| Sponsor: Zar | mbon S.p.A. | Protocol Number: | Z7224L02 |
|--------------|-------------|------------------|----------|
|--------------|-------------|------------------|----------|

# ZAMBON S.p.A

# STATISTICAL ANALYSIS PLAN

Protocol: Z7224L02

**EudraCT Number** 2016-004558-13

IND Number 134361

**Treatment: Inhaled Colistimethate Sodium** 

A DOUBLE-BLIND, PLACEBO-CONTROLLED, MULTI-CENTRE, CLINICAL TRIAL TO INVESTIGATE THE EFFICACY AND SAFETY OF 12 MONTHS OF THERAPY WITH INHALED COLISTIMETHATE SODIUM IN THE TREATMENT OF SUBJECTS WITH NON-CYSTIC FIBROSIS BRONCHIECTASIS CHRONICALLY INFECTED WITH PSEUDOMONAS AERUGINOSA (P. AERUGINOSA)

Author(s): PPD and PPD

Document Status: Version 4 FINAL

Version Dates: 8 April 2022

Pages: 92

#### STATEMENT OF CONFIDENTIALITY

This document is Zambon's sole property and ownership. This document, and all information and data contained herein has to be considered and treated as strictly confidential. This document shall be used only for the purpose of the disclosure herein provided. No disclosure or publication shall be made without the prior written consent of Zambon.

| Sponsor: | Zambon S.p.A. | Protocol Number: | Z7224L02 |
|----------|---------------|------------------|----------|
|----------|---------------|------------------|----------|

### APPROVAL PAGE

**Protocol Title:** A double-blind, placebo-controlled, multi-centre, clinical trial to investigate the efficacy and safety of 12 months of therapy with inhaled colistimethate sodium in the treatment of subjects with non-cystic fibrosis bronchiectasis chronically infected with *Pseudomonas aeruginosa* (*P. aeruginosa*)

**Protocol Name: Promis II** 

Protocol Code: Z7224L02

Protocol Version and Date: Version 5.0; 22 July 2021

**EudraCT number: 2016-004558-13** 

**IND number: 134361** 

Authors: PPD and PPD

Sponsor Name and Address: Zambon S.p.A.

Via Lillo del Duca 10

20091 Bresso - Milan - Italy

As agreed and approved by:



# **Contents**

Sponsor:

| A | BBRF | CVIATIONS | 6 |
|---|------------|-------------------------------------------------------|----|
| 1 | IN | TRODUCTION | 8 |
| 2 | ST | UDY OBJECTIVES | 9 |
| | 2.1 | Primary Endpoint | g |
| | 2.2 | SECONDARY ENDPOINTS | |
| | 2.3 | SAFETY ENDPOINTS | |
| 3 | | UDY DESIGN | |
| , | | | |
| | 3.1 | DISCUSSION OF STUDY DESIGN | |
| | 3.2 | STUDY TREATMENT | |
| | 3.3 | STUDY SCHEDULE | |
| | 3.3 | | |
| | 3.4 | .2 Trial Flow Chart - France | |
| | | CONCOMITANT MEDICATION | |
| | 3.5 | STUDY ANALYSIS POPULATIONS | |
| | | <u>-</u> | |
| | 3.5 | J I | |
| | 3.5 | J J 1 | |
| | 3.5 | 1 | |
| | 3.6 | 5.5 Other Populations Defined for Tables and Listings | |
| | | WITHDRAWN SUBJECTS | |
| | 3.7 | RANDOMISATION | |
| | 3.8<br>3.9 | BLINDING | |
| | | SAMPLE SIZE | |
| 4 | ST | ATISTICAL METHODOLOGY | 21 |
| | 4.1 | PLANNED ANALYSES | 21 |
| | 4.1 | .1 Populations for the Analysis | 21 |
| | 4.1 | .2 Treatment Groups | 22 |
| | 4.1 | 4 | |
| | 4.1 | .4 Statistical Significance | 22 |
| | 4.1 | .5 Subgroup Analyses | 22 |
| | 4.1 | .6 Definition of Baseline | 23 |
| | 4.1 | .7 Definition of Exposure Time and Follow-up Time | 23 |
| | 4.1 | .8 Visit dates | 24 |
| | 4.1 | .9 Date of First/Last IMP Dose | 24 |
| | 4.1 | .10 Data Re-Allocation | 24 |
| | 4.1 | .11 Exclusion of Data from the Statistical Analysis | 25 |
| | 4.1 | .12 Listings | 25 |
| | 4.2 | Interim Analysis | 25 |
| | 4.2 | .1 COI Committee | 25 |
| | 4.3 | DISPOSITION OF SUBJECTS | 26 |
| | 4.4 | BASELINE AND DEMOGRAPHIC CHARACTERISTICS | 26 |
| | 4.4 | .1 Demography Characteristics | 26 |
| | 4.4 | .2 Smoking and Alcohol Status | |

| Sporisor. | Zambon S.p.A. | Protocol Number. | Z1224L02 | |
|---|---|---|---|---|
| 4.4.3 | Non-CF Bronchiectasis Histo | orv | | 27 |
| | Past or Concomitant Relevan | • | | |
| | Spirometry at Visit 1 and Pre- | | | |
| | Haematology, Clinical Chemi | | | |
| | Vital Signs at Visit 1 | • | | |
| | Physical Examination at Visit | | | |
| | 12-Lead ECG at Visit 1 | | | |
| | Pregnancy Test | | | |
| | Presence of CCI | | | |
| | CCI and CCI | | | |
| | POSURE | | | |
| | Number and Duration of Inh | | | |
| | Exposure Days | | | |
| 4.5.3 | Extent of Exposure | | | 30 |
| 4.5.4 | Adherence | | | 30 |
| 4.5.5 | IMP interruptions | | | <i>31</i> |
| 4.6 Pri | IOR AND CONCOMITANT MEDIC | CATION | | 31 |
| 4.7 Eff | FICACY / PRIMARY AND SECON | DARY ANALYSIS | | 32 |
| 4.7.1 | Primary Endpoint | | | 32 |
| <b>4.7.2</b> 1 | Normality Assumption Check | ing | | 32 |
| 4.7.3 | Closed Testing Procedure for | Primary Analysis | | 32 |
| | Method of Analysis for Prima | | | 32 |
| 4.7.4. | 1 CCI Analysis Usin | | | |
| 4.7.4. | | _ | | |
| 4.7.4. | | | | |
| | Secondary Endpoint Analysis | | | |
| <b>4.7.6</b> 1 | Methods of Analysis for Seco | ndary Endpoints | | 38 |
| CCI | | | | |
| | | | | 44 |
| | FETY ANALYSIS | | | |
| | Adverse Events | | | |
| 4.8.1. | | | | |
| | Spirometry Results | | | |
| | CCI | | | 48 |
| | Haematology, Clinical Chemi | | | |
| | Vital Signs | | | |
| | Physical Examination Results | | | |
| | 12-Lead ECG | | | |
| 4.8.8 I | Pregnancy Test | | | 51 |

| Sponsor: | Zambon S.p.A. | Protocol Number: | Z7224L02 |
|---|---|---|---|
| 4.8.9 | Other Data | | 51 |
| | DJUSTMENT FOR COVARIATES | | |
| 4.9.1 | Country Effects | , | 52 |
| | OTOCOL DEVIATIONS | | |
| 4.10.1 | Major Protocol Deviation Cri | iteria | 52 |
| 4.10.2 | Protocol Deviations | | 53 |
| | ISSING DATA | | |
| 4.12 Di | EVIATIONS FROM THE SAP | | 55 |
| | HANGES IN CONDUCT OR PLANS | | |
| 4.14 A | LGORITHMS/SAS CODES | | 57 |
| 5 TABL | ES AND LISTINGS | | 65 |
| 5.1 TA | ABLE FORMAT | | 65 |
| Header | s | | 65 |
| Display | Titles | | 66 |
| 5.2 Co | ONVENTIONS | | 66 |
| 5.3 TA | ABLES | | 68 |
| | Section 14.1: Demographic a | | |
| | Section 14.2: Primary | | |
| | Section 14.2: Secondary | | |
| | Section 14.3: Safety | | |
| | STINGS | | |
| | GURES | | |
| 5.6 Ri | EFERENCES | | 74 |
| APPENDIX | (1: <mark>cc</mark> | CCI | 75 |
| APPENDIX | C2: CCI CCI | E CCI | 81 |
| APPENDIX | 3: WHO-DD PREFERRED | TERMS FOR ANTI | BIOTICS AND ANTI- |

| Sponsor: Zambon S. | A. Protocol Number: | Z7224L02 |
|--------------------|---------------------|----------|
|--------------------|---------------------|----------|

# **Abbreviations**

| CCI | CCI |
|------------------|-------------------------------------------------|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| ANCOVA | Analysis of Covariance |
| ATC | Anatomical Therapeutic Chemical |
| BMI | Body Mass Index |
| CA | Competent Authority |
| CF | Cystic Fibrosis |
| CFU | Colony Forming Units |
| CI | Confidence Interval |
| CRO | Contract Research Organisation |
| CS | Clinically Significant |
| CT | Computerised Tomography |
| CTP | Clinical Trial Protocol |
| CTR | Clinical Trial Report |
| CCI | Data CCI |
| EC | Ethics Committee |
| eCRF | electronic Case Report Form |
| eCOA | electronic Clinical Outcome Assessment |
| ED | Exposure Day |
| FEV <sub>1</sub> | Forced Expiratory Volume in one second |
| FOE | Frequency of Exacerbations |
| FVC | Forced Vital Capacity |
| GLI | Global Lung Function Initiative |
| ICH | International Conference on Harmonisation |
| IMP | Investigational Medicinal Product |
| ITT | Intention-To-Treat |
| IWRS | Interactive Web Response System |
| MAR | Missing At Random |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MI | Multiple Imputation |
| mITT | Modified Intention-To-Treat (Full Analysis Set) |
| MIU | Million International Unit |
| NCFB | Non-CF-Bronchiectasis |
| NCS | Non Clinically Significant |
| P. aeruginosa | Pseudomonas aeruginosa |
| PP | Per-Protocol |
| PT | Preferred Term |
| PWP | Prentice, Williams and Peterson |
| CCI | CCI |
| CCI | CCI |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |

| Sponsor. | Zambon S.p.A. | Protocol Number. | 2/224L02 |
|---|---|---|---|
| SD | Standard Deviation | | |
| CCI | | | |
| SOC | OC System Organ Class | | |
| SUSAR | Suspected Unexpected | Serious Adverse React | ion |
| TEAE | AE Treatment Emergent Adverse Event | | |
| WHO | HO World Health Organisation | | |

| Sponsor: Zambon S.p.A. Protocol Number: Z7224 | L02 |
|-----------------------------------------------|-----|
|-----------------------------------------------|-----|

# 1 Introduction

This document presents the Statistical Analysis Plan (SAP) for Zambon, Protocol No. Z7224L02: A double-blind, placebo-controlled, multi-centre, clinical trial to investigate the efficacy and safety of 12 months of therapy with inhaled colistimethate sodium in the treatment of subjects with non-cystic fibrosis bronchiectasis chronically infected with *Pseudomonas aeruginosa* (*P. aeruginosa*)

This analysis plan is based on the final protocol Version 5.0 dated 22Jul2021.

The SAP provides the description of the analysis for the final analyses. Any deviations from the SAP which occur after breaking the blind will be documented and justified in the final clinical trial report (CTR) and deviations will be clearly marked as 'post hoc' analysis.

| Sponsor: Zambon S.p.A. Protocol Number: Z7224L02 |
|--------------------------------------------------|
|--------------------------------------------------|

# 2 Study Objectives

The primary objective of the trial is to investigate the effect of the use of inhaled colistimethate sodium, administered twice daily via the collection for 12 months, compared to placebo in subjects with non-cystic fibrosis bronchiectasis (NCFB) chronically infected with *P. aeruginosa* on the annualized frequency of pulmonary exacerbations.

# 2.1 Primary Endpoint

The primary endpoint of this trial is the mean annual NCFB pulmonary exacerbation rate.

A pulmonary exacerbation is defined as the presence concurrently of at least 3 of the following 8 symptoms/signs for at least 24 hours:

- Increased cough;
- Increased sputum volume and/or consistency;
- Increased sputum purulence;
- New or increased haemoptysis;
- Increased wheezing;
- Increased dyspnoea;
- Increased fatigue/malaise;
- Episodes of fever (temperature ≥38°C);

And it is clinically determined that the subject requires and is prescribed systemic antibiotic therapy.

The start date of a protocol-defined pulmonary exacerbation will be taken as the first day that at least 3 of the pre-defined 8 symptoms/signs occurred concurrently for at least 24 hours, as determined by the Investigator, as documented by the start date of the corresponding AE in the eCRF AE form.

Resolution of a pulmonary exacerbation is defined as the date of completion of the required course(s) of systemic antibiotic treatment and/or the Investigator's judgement that the NCFB pulmonary exacerbation has resolved, as documented by the end date provided for the corresponding AE in the eCRF AE form, whichever is the later of the two dates. The exacerbation end date will be reported at the next scheduled visit or by phone. A new pulmonary exacerbation is only considered to occur if there are at least 14 days between the end of the course of systemic antibiotics and the onset of new qualifying symptoms.

Any episodes of pneumonia during the trial should be considered as pulmonary exacerbations. Episodes of pneumonia which are radiologically confirmed and/or requiring intravenous antibiotics and/or hospitalisation will be considered as severe pulmonary exacerbations. Adverse Events of COVID-19 with symptoms of an exacerbation, requiring antibiotics during the course of the study are considered as pulmonary exacerbations. All pulmonary exacerbations must have the associated

| Sponsor: Zambon S.p.A. | Protocol Number: | Z7224L02 |
|------------------------|------------------|----------|
|------------------------|------------------|----------|

Pulmonary Exacerbation, Pulmonary Exacerbation Symptoms and Systemic Antibiotic Therapy forms entered into the eCRF, and linked to the corresponding AE.

The treatment of pulmonary exacerbations will follow current treatment regimens used at the respective participating investigational site.

A supportive analysis will be conducted using an alternative definition of NCFB pulmonary exacerbation. The re-classification of exacerbations will be done in a blinded fashion (before database lock). Alternative definition of pulmonary exacerbation: deterioration in three or more of the following key symptoms for at least 48 hours:

- Cough;
- Sputum volume and/or consistency;
- Sputum purulence;
- Breathlessness and/or exercise tolerance (dyspnoea);
- Fatigue and/or malaise;
- · Haemoptysis;

And a physician determines a change in bronchiectasis treatment is required when other potential causes of clinical deterioration have been discounted.

# 2.2 Secondary Endpoints

The secondary endpoints of this trial are:



| Sponsor: | Zambon S.p.A. | Protocol Number: | Z7224L02 |
|----------|---------------|------------------|----------|



# 2.3 Safety Endpoints

The safety endpoints of this trial are:

- (1) Incidence of treatment emergent adverse events (TEAEs);
- (2) Absolute changes in percent-predicted forced expiratory volume in 1 second (FEV<sub>1</sub>) from baseline to each post-baseline visit;
- (3) The number of subjects experiencing bronchospasm clinically or spirometrically determined following IMP administration;
- from Screening/Randomisation (Visit 1/Visit 2) to Visits 3, 5 and end of treatment (Visit 7) as well as on confirmation (Visit 1/Visit 2) to Visits 3, 5 and end of treatment (Visit 7) as well as on confirmation (Visit 1/Visit 2) to Visits 3, 5 and end of treatment (Visit 7) as well as on confirmation (Visit 1/Visit 2) to Visits 3, 5 and end of treatment (Visit 7) as well as on confirmation (Visit 1/Visit 2) to Visits 3, 5 and end of treatment (Visit 7) as well as on confirmation (Visit 1/Visit 2) to Visits 3, 5 and end of treatment (Visit 7) as well as on confirmation (Visit 1/Visit 2) to Visits 3, 5 and end of treatment (Visit 7) as well as on confirmation (Visit 1/Visit 2) to Visits 3, 5 and end of treatment (Visit 7) as well as on confirmation (Visit 1/Visit 2) to Visits and clinic visits due to pneumonia;
- (5) CCI from Screening (Visit 1) to End of Treatment (Visit 7);
- (6) Haematology, clinical chemistry and renal function tests;
- (7) Physical examination and vital signs data;
- (8) 12-lead electrocardiogram.

| Sponsor: Zambon S.p.A. Protoco | Number: Z7224L02 |
|--------------------------------|------------------|
|--------------------------------|------------------|

# 3 Study Design

# 3.1 Discussion of Study Design

This is a randomised, multi-centre, double-blind, placebo-controlled, parallel-group interventional trial in subjects with NCFB suffering from chronic infections with *P. aeruginosa*.

The trial will be conducted in approximately 80 sites in up to 6 countries. A total of 420 subjects (210 in each treatment group) are planned to be enrolled into the trial. The enrolment is competitive among sites.

At Visit 2 (within 30 days after Visit 1), eligible subjects with *P. aeruginosa* cultured from an initial sputum sample will be randomised in a 1:1 ratio to receive either colistimethate sodium or placebo.

It is planned that subjects will be contacted by phone 7 days after Randomisation (Visit 2) to determine if there are any issues with IMP administration and/or any initial AEs and will, thereafter, attend 5 further visits at the sites at 1, 3, 6, 9, and 12 months after Randomisation (i.e. Visits 3, 4, 5, 6, and 7) and will have 1 follow-up phone call at 12.5 months. Additional clinic visits, where feasible, and weekly phone calls will be conducted following pulmonary exacerbations until resolution.

The maximum expected duration of participation in the trial for an individual subject, from Visit 1 (Screening) to the follow-up phone call is up to 13.5 months. Treatment duration will be 12 months.

The start of the trial is defined as first subject in, i.e. Visit 1 for the first subject. The end of the trial is defined as the last subject out, i.e. when the last subject has the follow-up phone call.

## 3.2 Study Treatment

At Visit 2 (within 30 days after Visit 1) eligible subjects with *P. aeruginosa* cultured from their initial sputum sample will be randomised in a 1:1 ratio to receive either colistimethate sodium or placebo.

Subjects will be administered the first dose of the IMP at the investigational site prepared by the site staff and will be instructed by the Investigator or a delegated person how to prepare and self-administer the IMP at home via the CCI Aerosol Delivery CCI system, twice daily (morning and evening) over a period of 12 months. Prior to each administration, a bronchodilator (salbutamol/albuterol) has to be taken.

Colistimethate sodium and placebo will be supplied in 30-vial packs.

Colistimethate sodium is supplied as sterile powder in a glass vial. Each vial contains 1,000,000 International Units (1 MIU) which weighs about 80 mg (equivalent to about 33 mg colistin base activity).

Identical sterile vials for placebo will be used. All vials will be masked with white plastic sleeves so that the contents are not visible. The weight of the powder is insignificant compared to the glass vial.

# 3.3 Study Schedule

The current trial will include 7 planned clinical visits at the investigational site, 1 telephone call 7 days after commencing treatment and 1 follow-up telephone call two weeks after discontinuation of treatment, as detailed in Section 9 of the CTP. A detailed flow chart of CTP Version 4.0 showing the procedures performed is given below in Table 3.3.1.

Additional procedures are scheduled for France sites according to CTP Version 4.0-FRA, as reported in Table 3.3.2.

| Sponsor: | Zambon S.p.A. | Protocol Number: | Z7224L02 |
|----------|---------------|------------------|----------|
|----------|---------------|------------------|----------|

### 3.3.1 Trial Flow Chart

| VISITS | Visit 1<br>Screening | Visit 2<br>Randomisation | Phone call | Visit 3 | Visit 4-6 | Visit 7<br>EoT | Follow-Up<br>'Phone Call | Exacer-<br>bation<br>Visit <sup>a</sup> |
|---|---|---|---|---|---|---|---|---|
| ACTIVITIES | Within 30 Days<br>of Visit 2 | Day 0 | Day 7 | Day 28<br>± 1 week | Every 3<br>months<br>± 1 week | 12 months<br>± 1 week | 2 weeks ± 3<br>days after<br>EoT | |
| Informed consent | X | | | | | | | |
| Medical history/demography | X | | | | | | | |
| Pregnancy test | X | X | | X | Х | X | | |
| Vital signs | X | | | | | X | | X |
| Physical examination | X | | | | | Х | | X |
| Previous/concomitant medications | X | X | | X | Х | Х | X | X |
| 12-lead ECG | X | | | | | Х | | |
| Obtain blood samples:<br>Haematology and clinical chemistry/Renal Function/PK* | х | Xc | | X <sup>a, c</sup> | X <sub>p</sub> | х | | |
| Collect sputum sample | Х | X | | X | X <sup>d</sup> | Х | | X |
| Verify eligibility for randomisation | Х | X | | | | | | |
| Spirometry: FEV <sub>1</sub> and FVC | X | Xe | | X | X | Xe | | X |
| CCI | | X | | X | Х | Х | | |
| Training, Dispensing/Collection | | X | | | | X | | |
| Review of IMP administration & column use (adherence) | | X | X | X | Х | Х | | |
| Study Medication: Dispense/Accountability | | X | | Х | Х | Х | | |
| Record of hospitalisations and days of work absence | | | Х | Х | Х | Х | | X |
| AE monitoring including exacerbations not otherwise reported | х | х | Х | Х | Х | Х | Х | X |
| Weekly follow up phone calls to determine end of Pulmonary Exacerbations | | | | | | | | X |

a; renal function test only. b; haematology, clinical chemistry and renal function test at Visit 5 (6 Months) only. c; PK sampling only (for relevant sites). d; Visit 5 only. e; FEV<sub>1</sub> and FVC to be measured pre-bronchodilator and 30 minutes post IMP dose.

| Sponsor: | Zambon S.p.A. | Protocol Number: | Z7224L02 |
|----------|---------------|------------------|----------|
|----------|---------------|------------------|----------|

# 3.3.2 Trial Flow Chart - France

| ACTIVITIES | Visit 1<br>Screening/<br>Rescreening | Visit 2<br>Randomisation | Phone call<br>1 week after<br>Visit 2 | Visit 3 | Visit 4 | Visit 5 | Visit 6 | Visit 7<br>End of<br>treatment <sup>c</sup> | Follow-up<br>phone call | Exacer-<br>bation<br>Visit <sup>a</sup> |
|---|---|---|---|---|---|---|---|---|---|---|
| | Day -30/-7 | Day 0 | Day 7 | Day 28<br>± 1 week | 3 months<br>± 1 week | 6 months<br>± 1 week | 9 months<br>± 1 week | 12 months<br>± 1 week | 2 weeks +/-<br>3 days after<br>EOT | |
| Informed consent | X | | | | | | | | | |
| Medical history/demography | X | | | | | | | | | |
| Inclusion/exclusion criteria | X | X | | | | | | | | |
| Check screen failure criteria | | X | | | | | | | | |
| Pregnancy test (urine dipstick) | X | X | | X | X | X | X | X | | |
| Vital signs | X | X | | X | X | X | X | X | | X |
| Physical examination (including chest auscultation) | X | | | | | | | Х | | X |
| Previous/concomitant medications<br>(including azithromycin/erythromycin use) | X | х | | X | Х | X | X | X | X | X |
| 12-lead ECG | X | | | | | | | X | | |
| Haematology and clinical chemistry | X | | | X <sup>d</sup> | X <sup>d</sup> | X | X <sup>d</sup> | X | | |
| Collect sputum sample | X | X | | X | | X | | X | | X |
| CCI | | X | | X | X | X | X | X | | |
| Spirometry: FEV <sub>1</sub> and FVC | X | Xb | | X | X | X | X | Xb | | X |
| Dispensing and training on CC | | X | | | | | | | | |
| collection <sup>c</sup> | | | | | | | | X | | |
| IMP administration under clinical supervision and training on IMP preparation | | Х | | | | | | X | | |
| Study Medication: dispensing | | X | | X | X | X | X | | | |

| Sponsor: | Zambon S | bon S.p.A. | | | Protocol Number: | | | 2 | Z7224L02 | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Check of any issue on the mand administration of IMP and to nebuliser device (adherence) | he use of the | | | х | | | | | | | | |
| Check on NCFB pulmonary | exacerbations | | X | | | X | X | X | X | X | | X |
| Record of hospitalisations an work absence | ıd days of | | | | | X | X | X | X | х | | X |
| Study Medication collection accountability | and vials | | | | | X | X | X | X | Х | | |
| AE monitoring | | X | X | X | | X | X | X | X | X | X | X |

a Exacerbation Visit may occur from Visit 2 to Visit 7 (the following has to be recorded: start date and duration of all symptoms, review of all symptoms, concomitant medications (including antibiotics), physical examinations and vital signs, spirometry [FEV1, FVC] if feasible, date of policy physical examinations are physical examinations.

b FEV<sub>1</sub> and FVC to be measured pre-salbutamol/albuterol and 30 minutes post IMP dose.

will be returned by subject, to download data on actual subject's compliance.

d Only renal function tests (creatinine and BUN) will be performed.

<sup>\*</sup> PK is handled separately and is outside the scope of this SAP.

| Sponsor: Zambon S.p.A. Protocol Number: Z7224L02 |
|--------------------------------------------------|
|--------------------------------------------------|

### 3.4 Concomitant Medication

Permitted concomitant medications are reported in Section 11 of the CTP.

## 3.5 Study Analysis Populations

There will be 4 analysis populations defined for the trial analyses:

### 3.5.1 Intention-To-Treat Population

The Intention-To-Treat Population (ITT) will include all subjects who provided informed consent and received a patient number (randomisation number) whether or not they receive IMP.

Following the ITT principle, subjects will be analysed according to the treatment they have been assigned to at randomisation.

### 3.5.2 Modified Intention-To-Treat Population

The modified ITT (mITT) Population will comprise all subjects who provided informed consent, were randomised and received at least 1 dose or partial dose of the IMP.

Subjects will be analysed according to the treatment they have been assigned to at randomisation.

The mITT will be used to produce summaries of baseline subject characteristics and for the analysis of all primary and secondary efficacy endpoints. Minimal difference in sample size is expected between ITT and mITT. Being a double-blind study, no bias due to the exclusion of the non-treated subjects is expected. Exposure variables will also be presented for the mITT.

### 3.5.3 Safety Population

The Safety Population will comprise all subjects who provided informed consent, were randomised and received at least 1 dose or partial dose of IMP.

Subjects will be analysed according to the treatment they actually received.

The Safety Population will be used to produce summaries of all safety related endpoints and demography.

#### 3.5.4 Per-Protocol Population

The Per-Protocol Population (PP) will include all mITT subjects who were considered compliant with study drug administration (i.e. had an adherence of at least 80%) and who had no major protocol deviations that were considered as potentially impacting the efficacy results.

Major protocol deviations might include, but are not limited to, subjects taking a not-permitted concomitant medication, the IMP not being administered during the trial as defined in the protocol, subjects receiving a treatment different than the one assigned by randomisation. Categories of protocol deviations and additional details are reported in Section 4.10. The exact definition of major protocol deviations impacting the efficacy results will be discussed by the study team during the blind review of the data and described in the Blind Data Review and Analysis Sets Report.

Results of the primary and relevant secondary efficacy endpoints analyses conducted for the

| Sponsor: Zambon S.p.A. | Protocol Number: | Z7224L02 |
|------------------------|------------------|----------|
|------------------------|------------------|----------|

PP will be considered as supportive.

### 3.5.5 Other Populations Defined for Tables and Listings

For the purposes of tables and listings, a further 3 populations are defined:

- All screened subjects: all subjects who provide informed consent;
- Screening failure subjects: all subjects who provide informed consent and are screening failures;
- Enrolled subjects: all subjects who provide informed consent and are not screening failures.

# 3.6 Withdrawn Subjects

Subjects will be withdrawn from the trial for one of the following reasons:

- subject may withdraw from the study at any time at his/her own request;
- subject may withdraw from the study due to an AE including subjects experiencing a
  decrease in FEV<sub>1</sub> >15% from pre-bronchodilator baseline and/or clinically determined
  bronchospasm after receiving their first dose of IMP;
- subject may be withdrawn at any time at the discretion of the Investigator for safety, behavioural, compliance or administrative reasons;
- subject may be withdrawn due to lack of adherence to study medication regimen;
- subjects who become pregnant should be withdrawn from the trial;
- lost to follow-up: before a subject is deemed lost to follow-up, the Investigator or designee must make every effort to regain contact with the participant (where possible, 3 telephone calls and, if necessary, a certified letter to the participant's last known mailing address or local equivalent methods). These contact attempts should be documented in the participant's medical record. Should the participant continue to be unreachable, he/she will be considered to have withdrawn from the study;
- Sponsor, CA, or EC/IRB(s) terminate the trial or participation of an individual site.

The reason for removal of a subject from the trial or premature discontinuation of treatment must be fully documented in the electronic case report form (eCRF) as well as in respective source documents.

Any subject who withdraws after randomisation will not be replaced. Withdrawn subjects will not be re-entered into the study.

## 3.7 Randomisation

At Visit 2, eligible subjects will be randomised using the interactive web response system (IWRS) according to a pre-specified randomisation scheme such that they either receive colistimethate sodium or placebo. Site and use of stable concomitant therapy with oral macrolides (e.g. azithromycin or erythromycin or clarithromycin) (Yes/No) will be considered as factors for balancing randomisation, i.e. stratification factors. Thus, within each site, subjects

with oral macrolides use will be randomised independently from subjects without use of macrolides, to receive colistimethate sodium or placebo in a 1:1 ratio. The randomisation within each site and nested level macrolide use will be done with blocks to guarantee a good balance between colistimethate sodium and placebo at any stage of the enrolment.

Note: according to Exclusion Criterion 15, the decision on whether stable concomitant antibiotic therapy with oral macrolides will be administered to a subject or not will have been taken at least 30 days prior to the Screening Visit (Visit 1). The treatment with oral macrolides should be continued throughout the trial in order not to jeopardize the study results.

# 3.8 Blinding

Investigational site staff including the Investigator and all personnel involved in study procedures will be blinded to treatment allocation. All Contract Research Organisation (CRO) and Zambon study staff involved in monitoring, data management, or other aspects of the study will also be blinded.

The allocation to treatment will be stored within the IWRS database until unblinding of the trial is requested.

The code for any individual subject will not be broken by the Investigator during the course of the trial except in the circumstance of a Serious Adverse Event (SAE) where knowledge of treatment assignment is essential for the management of patient care. CRO and Zambon Pharmacovigilance can unblind subjects in case of suspected unexpected serious adverse reactions (SUSARs) to be reported to the competent authority (CA) and ethics committees (ECs).

The randomisation code will be provided to the Biostatistics group once written authorization of database lock has been received and analysis populations have been defined.

# 3.9 Sample Size

Under these assumptions, CCI



CONFIDENTIAL

exacerbation (FOE), with a two-sided significance level of color, a treatment effect of color and a follow-up time of 1 year, assuming a frequency of color pulmonary exacerbations per annum

allowing for over-dispersion for frequency of

| Sponsor: Zambon S.p.A. | Protocol Number: | Z7224L02 |
|------------------------|------------------|----------|
|------------------------|------------------|----------|

for the FOE, a sample size of 170 completed subjects per group will provide a power of 90% (simulated in street size). If the treatment effect size is collaboration between the collistimethate sodium and placebo groups, the power with coll completed patients per group will be coll.

Assuming a drop-out rate of about 20%, the total sample size should be 210 subjects per treatment group (420 total subjects).

In November 2021, recruitment to PROMIS II was stopped based on the very positive data from PROMIS I, giving rise to ethical concerns of continuing to expose subjects to placebo in PROMIS II, the potential loss of scientific equipoise in the context of the PROMIS I results, and PROMIS II being unable to complete in a reasonable time frame, primarily related to the COVID-19 pandemic.

At the time that recruitment into PROMIS II was stopped, 287 of the originally planned 420 had been randomised. All subjects will be brought back for Visit 7 or an early termination visit on or before the end of February 2022.

| Sponsor: | Zambon S.p.A. | Protocol Number: | Z7224L02 |
|----------|---------------|------------------|----------|
| • | - | | |

# 4 Statistical Methodology

# 4.1 Planned Analyses

The statistical analysis will be performed by CCI and will be carried out according to International Conference on Harmonisation (ICH) guidelines ICH E9: "Statistical Principles for Clinical Trials" (CPMP/ICH/363/96 September 1998) and ICH E10 "Choice of Control Group in Clinical Trials" (CPMP/ICH/364/96 January 2001).

All the statistical analyses and outputs will be produced using SAS release 9.4 or later (SAS Institute, Inc. Cary, NC, USA).

The data from all countries and all sites will be pooled and summarised. Unless stated otherwise, all available data from withdrawn subjects will be included in the analysis up to the time of withdrawal.

### 4.1.1 Populations for the Analysis

Demographics and baseline characteristics will be summarised for the mITT population. Demographics and selected baseline characteristics will be also presented for the Safety Population.

The following baseline characteristics will be presented on the mITT Population only:

- Smoking and Alcohol Status
- Non-CF Bronchiectasis History
- Past and Concomitant Relevant Diseases, Diagnosis or Surgeries
- Prior and Concomitant Medication.

No baseline testing will be performed.

Primary and relevant secondary efficacy variables will be summarised and analysed for the mITT and PP Population. Results on PP will be considered as supportive. CCI will only be done on the mITT population.

The number of days of work absence and hospitalisations will be analysed for the mITT population only.

The exposure data will be analysed on the Safety and mITT Populations.

The safety variables will be summarised for the Safety Population.

In case an error occurs in treatment allocation, the following rules will be followed:

- If a subject was randomised but received the incorrect treatment for all the time the subject
  was in the study, he/she will be reported under the randomised treatment group for all
  analyses performed on the ITT and on the mITT Population (and in listings on all screened
  subjects). He/she will be reported under the treatment actually received for all analyses
  performed on the Safety Population (i.e. an as-treated analysis will be performed). Such
  subjects will be excluded from the PP Population.
- If a subject received the incorrect treatment after being treated with the correct one, it's
  foreseen that the subject will be withdrawn from the study. Data for this subject will be

| Sponsor: | Zambon S.p.A. | Protocol Number: | Z7224L02 |
|----------|---------------|------------------|----------|
|----------|---------------|------------------|----------|

analysed until the date of the wrong treatment dispensing. All the data collected after that date will be reported in listings and flagged, but not included in the summary statistics. He/she will be reported under the randomised treatment group for all analyses performed and listings presented.

### 4.1.2 Treatment Groups

Statistics will be displayed for the following treatment groups:

- Colistimethate Sodium
- Placebo
- Overall.

### 4.1.3 Descriptive Statistics

Descriptive statistics will be used to summarise all efficacy and safety results.

Descriptive statistics for quantitative variables will include n (the number of observations, i.e. non-missing values), mean, standard deviation (SD), median, minimum and maximum values. The 25<sup>th</sup> and 75<sup>th</sup> percentiles will also be presented where clearly stated.

Categorical variables will be summarised by using frequency count and percent distributions. Percentages will be calculated using the total number of subjects per treatment/population.

### 4.1.4 Statistical Significance

The analysis of the trial is on a comparative basis. For all efficacy parameters, comparisons will be made between colistimethate sodium and placebo. Two-sided p-values <0.05 will be considered statistically significant and 95% two-sided confidence intervals (CIs) will be presented where appropriate. A hierarchical testing procedure will be applied to the secondary endpoints as detailed in Section 4.7.5 to maintain Type I Error control.

### 4.1.5 Subgroup Analyses

The mean annual NCFB pulmonary exacerbation rate will also be estimated in the following subgroups:

1. Number of NCFB pulmonary exacerbations requiring oral or intravenous antibiotics in the 12 months prior to study entry.

The number of NCFB pulmonary exacerbations requiring oral antibiotics in the last 12 months and the number of NCFB pulmonary exacerbations requiring intravenous antibiotics in the last 12 months prior to study entry, as collected in the eCRF Screening folder on the Non-CF Bronchiectasis History form, will be summed.

Subgroup results will be presented for subjects with 1, 2 and >2 NCFB pulmonary exacerbations in the last 12 months.

Subjects with no data regarding the number of NCFB pulmonary exacerbations requiring oral and/or intravenous antibiotics in the last 12 months prior to study entry will be excluded from the analysis.

| Sponsor: | Zambon S.p.A. | Protocol Number: | Z7224L02 |
|----------|---------------|------------------|----------|
|----------|---------------|------------------|----------|

2. Previous usage of colistimethate sodium/colistin (as collected on the Non-CF Bronchiectasis History eCRF form).

Based on data collected on the Non-CF Bronchiectasis History eCRF form regarding previous usage of Colistimethate Sodium/colistin, the subjects will be classified into one of the following groups:

- i. Without any previous usage of colistimethate sodium/colistin;
- ii. With previous usage of colistimethate sodium/colistin.

Subjects with missing data regarding previous usage of colistimethate sodium/colistin will be excluded from the analysis.

will be presented classifying subjects by status of previous usage of colistimethate sodium/colistin as collected on the Non-CF Bronchiectasis History eCRF form. Subjects with missing data regarding previous usage of colistimethate sodium/colistin will be included in the analysis in a separate 'unknown' subgroup.

Additional subgroup analyses for the mean annual NCFB pulmonary exacerbation rate endpoint will include:

- 4. Age at Visit 1 (<65, >=65)
- 5. Sex (Female, Male)
- 6. Country; for this, and all analyses using country, the small countries with few subjects will be grouped into a single 'Other' country category. Based upon blinded data, the smaller countries to be grouped are: Germany (N=3), Greece (N=3), Israel (N=4), Italy (N=1), New Zealand (N=6) and Portugal (N=2)
- 7. Adherence (compliance to IMP <80%, >=80%, Unknown).

### 4.1.6 Definition of Baseline

Age, height, weight and Body Mass Index (BMI) recorded at Visit 1 will be presented as baseline characteristics.

For 12-lead ECG, vital signs, physical examination and haematology, clinical chemistry and renal function parameters, baseline values are those recorded at Screening (Visit 1). If no assessment has been conducted at that visit, the last available value before IMP first dose (collected during unscheduled visits before IMP first dose) will be considered as baseline.

For sputum analysis, CCI and and spirometry baseline values are those recorded at Visit 2 before IMP first dose. If no assessment has been conducted at that visit, the last available value before IMP first dose (collected at the Screening visit or unscheduled visits before IMP first dose) will be considered as baseline.

### 4.1.7 Definition of Exposure Time and Follow-up Time

All the efficacy analyses are focused on the endpoints collected during the treatment period. For these analyses, the exposure time will not include the time from end of treatment to the follow-up call.

The exposure time in days will be calculated using the following formula:

| Sponsor: | Zambon S.p.A. | Protocol Number: | Z7224L02 |
|----------|---------------|------------------|----------|

 Exposure time (days) = [date of treatment completion/discontinuation - date of first IMP dose + 1].

The exposure time in years will be calculated using the following formula:

• Exposure time (years) = Exposure time (days) / 365.25.

Date of treatment completion will be the date of End of Treatment Visit.

Date of treatment discontinuation will be the date of End of Study Visit for subjects who discontinued the study before the End of Treatment Visit. In case a subject is lost to follow-up, the date of treatment discontinuation will be the date of last Study Visit.

Date of last exposure will not include any visits/calls after the end of treatment.

The follow-up time in days will be calculated using the following formula:

Follow-up time (days) = [date of study completion/discontinuation - date of first IMP dose + 1].

The follow-up time in years will be calculated using the following formula:

• Follow-up time (years) = Follow-up time (days) / 365.25.

#### 4.1.8 Visit dates

For each visit, the date recorded by the Investigator in the eCRF (variable SVSTDTC in the SDTM SV domain) will be considered as the visit date in all the algorithms and the listings.

#### 4.1.9 Date of First/Last IMP Dose

The date of first IMP dose is the earliest date of IMP dose considering both the eCRF and the recordings from the collision logging system.

The date of last IMP dose is derived as follows. Where data is available for the subject, the date of last IMP dose will be defined as the latest date from the logging system, with the following exception. Due to the Covid-19 pandemic, for some subjects, Visit 7 was split into a remote phone call (at the scheduled time of treatment completion), followed by an inclinic visit (for the purpose of collecting pre-dose and post-dose spirometry data to test for bronchospasm). In such cases, the scheduled study treatment period was completed at the time of the remote Visit 7 phone call, but an additional IMP dose was given at the time of the inclinic Visit 7. In these circumstances, the latest date from the logging system will be compared to the penultimate date from the logging system and, if the latest date is more than 14 days after the penultimate date (latest date – penultimate date >14), the logging system data will be used taking into consideration the penultimate IMP dose as the date of last IMP dose. The date of last IMP dose will be defined as the date of last IMP administration as entered on the End of Study eCRF form only when logging data is unavailable.

Any inconsistency between eCRF and coll logging system data will be discussed before the database lock.

### 4.1.10 Data Re-Allocation

Data collected at the early termination visit (when used) for discontinued subjects will not be re-allocated. Early termination data will not be moved in the database, however, statistical

programming will allocate this visit as Visit 7 within the Analysis Data Model (ADaM) datasets.

Potential issues of the approach defined above and other decisions regarding data re-allocation will be evaluated during the blind review of the data and documented in the Blind Data Review and Analysis Sets Report.

### 4.1.11 Exclusion of Data from the Statistical Analysis

If a subject received the incorrect treatment after being treated with the correct one, all the data collected after the date of the wrong treatment dispensing will be reported in listings and flagged, but not included in the statistical analysis on the ITT, mITT, Safety and PP populations.

Unless stated otherwise, primary efficacy endpoint and related assessments conducted at an early termination visit or unscheduled visit will be included in the statistical analysis, Where not stated differently, other assessments conducted at an early termination visit and unscheduled assessments will not be considered in the statistical analysis, but will be listed only.

Only NCFB pulmonary exacerbations with a start date  $\geq$  date of first IMP dose and  $\leq$  date of treatment completion/discontinuation will be considered in the analysis.

In case of data excluded from the statistical analysis (in the situations described above but also in other cases, for example: spirometry tests excluded due to technical issues, or assessment not done), the derived variables based on these data will not be calculated. For example, the change from baseline to Visit 5 will not be calculated if the measurement at Visit 5 is excluded from the statistical analysis, or all the changes from baseline will not be calculated if the measurements pre-dose are excluded.

### 4.1.12 Listings

All data collected will be presented in the listings.

# 4.2 Interim Analysis

No interim analysis is planned for this study. The trial terminated early, see Section 3.9.

# 4.2.1 Data CC

Committee Collecto evaluate the impact of decisions made on the integrity of the study data. Although the Collection will only review blinded data, the Collection will advise if additional collection analyses may be needed as a result of this pandemic. In addition, the Collection will review blinded pulmonary exacerbation data to determine whether or not events have been correctly assigned as meeting protocol-defined criteria. The Collection may recommend that sites reconsider their classification of pulmonary exacerbations as meeting the protocol-defined criteria or not (as well as re-examine the duration of the event based on the existing eCRF data), however, the ultimate decision will remain that of the Principal Investigator at each site.

Due to the impact of Covid-19 during the conduct of the study, the Sponsor has established a

| Sponsor: Zambon S.p.A. Protocol Number: Z7224 | L02 |
|-----------------------------------------------|-----|
|-----------------------------------------------|-----|

## 4.3 Disposition of Subjects

The number of subjects screened and the number of screen failures will be presented (overall). All screened subjects will be included. Re-screened subjects will be counted twice in the number of screened subjects. The number of re-screened subjects will be presented.

The number and percentage of randomised subjects who completed the study, withdrew from the study after randomisation and the number and percentage of subjects with each reason for withdrawal from the study will be presented by treatment group for the ITT population. Summaries of enrolled subjects will be reported overall and by country. These will include a presentation of country, number of subjects randomised and number of subjects who completed the study for the ITT population.

The number and percentage of subjects at Visit 2, who attended Visits 3, 4, 5, 6 and 7 and who had a follow-up call will be presented by treatment group and overall for the mITT Population. Time to completion/discontinuation from the study (days) will be summarised by descriptive statistics and calculated as (date of completion/discontinuation – date of first IMP dose).

The number and percentage of screened subjects who had any inclusion/exclusion criteria deviation as detailed in the eCRF will be reported. Results will be presented also for each criterion.

Protocol deviations affecting the efficacy analyses and protocol deviations specifically related to the COVID-19 pandemic will also be summarised for the Enrolled Population. The number and percentage of subjects included in each analysis population will be presented overall and by treatment group.

# 4.4 Baseline and Demographic Characteristics

No formal comparison between treatment groups on baseline and demographic characteristics will be done. Unless specifically stated in the relevant section, analysis will be done on the mITT Population.

### 4.4.1 Demography Characteristics

Demographics will be summarised by treatment group and overall. This will include age, ethnicity, gender, race, employment status, height (cm), weight (kg), BMI (kg/m²).

Summaries will be produced using the mITT and the Safety Population.

#### Note:

Age, height, weight, BMI and employment status recorded at Visit 1 will be presented.

## 4.4.2 Smoking and Alcohol Status

Smoking status at Screening (non-smoker, former smoker or current smoker), will be presented by treatment group and overall for the mITT Population. Former smoker will be further characterised summarising time from last cigarette (years) and number of pack-years.

Alcohol Status (Alcohol consumer: Yes or No) at Screening will be presented by treatment group and overall, along with summaries of alcohol units per week for alcohol consumers.

| Sponsor: Zambon S.p.A. | Protocol Number: | Z7224L02 |
|------------------------|------------------|----------|
|------------------------|------------------|----------|

#### Notes:

- For former smokers, time from last cigarette (years) will be calculated as (screening date date of last cigarette)/365.25;
- In order to calculate the time from last cigarette, the following rules will be applied for partial dates of the last date of smoking:
  - if only the day is missing, the first day of the month will be assumed;
  - if the day and the month are missing, then the first day of the year will be assumed.

### 4.4.3 Non-CF Bronchiectasis History

The following variables will be summarised for the mITT Population by treatment group and overall:

- Time since diagnosis of non-CF bronchiectasis (years);
- Diagnostic technique used (computerised tomography [CT] or high resolution CT: Yes or No);
- Number of lobes affected (1, 2, 3, more than 3);
- Underlying cause of the bronchiectasis;
- Number of NCFB pulmonary exacerbations requiring oral antibiotics in the last 12 months before Screening;
- Number of NCFB pulmonary exacerbations requiring intravenous antibiotics in the last 12 months before Screening;
- Previous usage of colistimethate sodium/colistin;
- Having at least 1 positive sputum culture for *P. aeruginosa* before Screening.

### Notes:

- Time since diagnosis of NCFB (years) will be calculated as (date of Visit 1 date of diagnosis of NCFB)/365.25;
- In order to calculate the time since diagnosis of NCFB, the following rules will be applied for partial dates of the date of diagnosis of NCFB:
  - if only the day is missing, the first day of the month will be assumed;
  - if the day and the month are missing, then the first day of the year will be assumed.

### 4.4.4 Past or Concomitant Relevant Diseases, Diagnoses or Surgeries

Past or concomitant relevant diseases, diagnosis or surgeries will be summarised by system organ class (SOC) and preferred term (PT), by treatment group and overall using the mITT Population.

#### Notes:

| Sponsor: | Zambon S.p.A. | Protocol Number: | Z7224L02 |
|----------|---------------|------------------|----------|
|----------|---------------|------------------|----------|

- Past or concomitant relevant Diseases, Diagnoses or Surgeries will be coded according to the Medical Dictionary for Regulatory Activities (MedDRA) version 19.1 or higher;
- Past relevant Diseases, Diagnoses or Surgeries are defined as records in the Medical History eCRF form which are not ongoing at Visit 1;
- Concomitant relevant Diseases, Diagnoses or Surgeries are defined as records in the Medical History eCRF form which are ongoing at Visit 1;
- Terms will be displayed in descending overall frequency (and then alphabetically) of SOCs and in descending overall frequency (and then alphabetically) of PTs within each SOC.

### 4.4.5 Spirometry at Visit 1 and Pre-Dose at Visit 2

The following spirometry parameters will be summarised by treatment group and overall:

- FEV<sub>1</sub> (L);
- Predicted FEV<sub>1</sub> (%);
- FVC (L);
- Predicted FVC (%).

Spirometry results assessed at Visit 1 and at Visit 2 Pre-dose will be summarised using summary statistics for continuous variables. Summaries will be provided for the mITT and for the Safety Population. Results for the Safety Population will be presented along with summaries for spirometry parameters assessed during Visits 3-7, inclusive.

More details of the analysis are reported in Section 4.8.2.

### 4.4.6 Haematology, Clinical Chemistry and Renal Function Parameters at Visit 1

Haematology, clinical chemistry and renal function parameters assessed at Visit 1 will be listed. More details of the analysis are reported in Section 4.8.4.

### 4.4.7 Vital Signs at Visit 1

Respiratory rate (breaths per minute), heart rate (beats per minute), systolic and diastolic blood pressure (mmHg) and body temperature (°C) assessed at Visit 1 will be listed.

More details of the analysis are reported in Section 4.8.5

### 4.4.8 Physical Examination at Visit 1

Physical Examination findings collected at Visit 1 will be listed.

More details of the analysis are reported in Section 4.8.6.

### 4.4.9 12-Lead ECG at Visit 1

The 12-lead ECG overall interpretation at Visit 1 will be listed.

More details of the analysis are reported in Section 4.8.7.

| Sponsor: Zambon S.p.A. | Protocol Number: | Z7224L02 |
|------------------------|------------------|----------|
|------------------------|------------------|----------|

### 4.4.10 Pregnancy Test

Results from the dipstick urine pregnancy test for women of child-bearing potential will be listed only.

### 4.4.11 Presence of Column at Visit 1

Number and percentage of subjects with presence of Collected at Visit 1 will be reported for the mITT Population. Subjects with results collected at Visit 2 will be considered as negative based on the central lab specifications. The local laboratory result will just record presence or absence of collected for eligibility purposes only. The number and percentage of subjects with presence of collected in the eCRF will be presented.

### 4.4.12 **CCI** and **CCI** B

The  $\square$  total score and domain scores and the  $\square$  domain scores at Visit 2 (see Sections 4.7.6.2 and 4.7.6.9 for further details regarding the calculation of the  $\square$  and  $\square$  will be summarised by treatment group and overall using the mITT Population and the PP Population for  $\square$  and the mITT Population only for  $\square$  (see Section 4.7.5). Results will be presented along with summaries for results at Visits 3 – 7, inclusive.

# 4.5 Exposure

#### 4.5.1 Number and Duration of Inhaled Doses

An inhaled dose is defined as any complete or partial dose of IMP that the subject inhaled either at the investigational site or at home (excluding doses ≤12.5% as recorded in the collapsing system and any final dose recorded in the collapsing system that is more than 14 days after the penultimate dose in the collapsing system where Visit 7 was split due to Covid-19, as described in Section ).

For doses administered at the investigational site, inhaled doses are all doses with a date of administration filled in the "IMP administration under clinical supervision" eCRF page. Complete doses are those recorded as complete in the eCRF. Partial doses are those recorded as non-complete in the eCRF.

For doses administered at home, inhaled doses are all doses with a date and time of administration recorded in the oclapsing system and dose different than "Null" or "\leq12.5%".

The overall number of inhaled doses either at the investigational site or at home will be summarised along with their duration. For doses administered at the investigational site only, the number of complete and partial doses will also be reported.

Summaries will be presented for the Safety and mITT Populations.

### Notes:

• All the doses will be recorded in the collaboration logging system, regardless of being administered at the investigational site or at home. Doses administered at home are those not recorded in the eCRF. In case of any inconsistencies between eCRF and collaborations.

data, the **local** data will be used in the analysis. While missing date/time of doses might be present in the eCRF, **coll** data are expected to be complete.

### 4.5.2 Exposure Days

An Exposure Day (ED) is defined as any day that the subject inhaled at least one full or partial dose of IMP as defined in Section , either at the investigational site or at home regardless of the number of doses on that day. The number of EDs per subject will be summarised overall and by treatment group for the Safety and mITT Populations using descriptive statistics for continuous variables.

### 4.5.3 Extent of Exposure

Extent of exposure (days) will be calculated using the following formula:

 Extent of exposure (days) = Date of last full or partial inhaled dose of IMP - date of first full or partial inhaled dose of IMP + 1.

The date of last full or partial inhaled dose of IMP is as defined in Section .

The extent of exposure will also be calculated in weeks using the following formula:

Extent of exposure (weeks) = Extent of exposure (days) / 7.

Dose of IMP either at the investigational site or at home will be considered.

Treatment exposure will be summarised overall and by treatment group for the Safety and mITT Populations using descriptive statistics for continuous variables.

### 4.5.4 Adherence

Adherence will be calculated overall.

The evaluation of adherence will be based on the following formula:

• Adherence (%) = (# Total Inhaled Doses / # Scheduled Doses)\*100.

The total number of inhaled doses of IMP will be computed as described in Section 4.5.1. In cases where, due to the Covid-19 pandemic, the final dose registered on the covid-19 device is the dose given at the in-clinic part of a split Visit 7 for the purposes of bronchospasm testing, any dose on the covid-19 that is later than the date of last IMP administration as entered on the End of Study eCRF form will not be counted as an inhaled dose for the calculation of IMP adherence.

The scheduled doses will be computed as 2 times the total number of days from Visit 2 to the end of period date, i.e. (End of period date – date of Visit 2) + 1.

For the overall adherence, the end of period date will be the date of the last inhaled dose of IMP, based on the latest of the last dose recorded in the column download (with the exceptions noted above relating to split Visit 7's) or the date of the last dose of IMP recorded in the End of Study form in the eCRF.

Adherence will be summarised by treatment group and overall for the mITT Population, presenting descriptive statistics for continuous variables and absolute and relative percentages of subjects considered to be adherent, i.e. with a least 80% of adherence.

| Sponsor: | Zambon S.p.A. | Protocol Number: | Z7224L02 |
|----------|---------------|------------------|----------|
|----------|---------------|------------------|----------|

An additional summary displaying the number and percentage of subjects in the following categories will also be presented by treatment group:

- < 60%;
- 60 to <70%:
- 70 to <80%;
- 80 to <90%;
- ≥90%.

## 4.5.5 IMP interruptions

The number and percentage of subjects with at least one IMP interruption, the number and percentage of subjects with at least one IMP interruption due to NCFB pulmonary exacerbation and the number of NCFB pulmonary exacerbations which lead to an IMP interruption will be presented.

Moreover, the number of days of IMP interruption overall and due to NCFB pulmonary exacerbations will be summarised using descriptive statistics for continuous variables.

Results will be presented overall and by treatment group for the Safety and mITT Populations.

#### Notes:

- NCFB pulmonary exacerbations will be linked to the corresponding AE using the AE number collected in the eCRF form "Pulmonary Exacerbation", i.e. "Please specify corresponding Adverse Event number for this Pulmonary Exacerbation".
- IMP interruption (days) will be calculated considering stop date and re-start date of IMP as collected in the eCRF "Adverse Event" form using the following formula:
  - IMP interruption (days) = Re-Start date of IMP date of Stop of IMP + 1.
- If any dose with a dose different than "Null" is recorded in the coll logging system during this period, then the coll data will be considered to compute IMP interruption: stop date will be the last IMP dose date before the start of the AE, re-start date will be the first IMP dose date after the start date of the AE.

### 4.6 Prior and Concomitant Medication

The incidence of prior and concomitant medications will be presented by therapeutic area according to the Anatomical Therapeutic Chemical (ATC) level 4 classification and preferred drug name, by treatment and overall for the mITT Population.

Prior medications are those that started and stopped before exposure to IMP; concomitant medications are all medications taken during the study period, including those started before but on going at first IMP dose.

Where a medication start/stop date is partially or fully missing, and it is unclear as to whether the medication is prior or concomitant, it will be assumed that it is concomitant.

#### Notes:

| Sponsor: | Zambon S.p.A. | Protocol Number: | Z7224L02 |
|----------|---------------|------------------|----------|
|----------|---------------|------------------|----------|

- Prior and concomitant medications are all medications collected in the eCRF forms
   Prior and Concomitant Medications and Systemic Antibiotic Therapy.
- Medications are coded using the World Health Organisation (WHO) Drug Dictionary, WHO-DD (please refer to the final Data Management Plan for the latest coding information);
- Only the number of subjects with medications (not the number of medications) will be presented;
- If a subject has multiple occurrences of a medication, the subject will be presented only
  once in the respective subject count;
- Prior and concomitant medications will be summarised in separate tables;
- Medications will be displayed in descending ATC text and drug name frequency overall and then alphabetically.

## 4.7 Efficacy / Primary and Secondary Analysis

The analysis of the trial is on a comparative basis. For all efficacy parameters, summaries will be presented by treatment group and comparisons will be made between colistimethate sodium versus placebo. Two-sided p-values <0.05 will be considered statistically significant and 95% two-sided CIs will be presented, where appropriate.

Primary and secondary efficacy variables, where not stated differently, will be summarised for the mITT and, where relevant, PP Populations. The primary analysis will be performed on the mITT Population. Analyses conducted using the PP will be considered supportive.

The health economic variables will be analysed on the mITT Population only.

### 4.7.1 Primary Endpoint

The primary endpoint of this trial is the annual NCFB pulmonary exacerbation rate.

The analysis of this endpoint requires for each subject both their count of NCFB pulmonary exacerbations and their exposure to randomised treatment. NCFB pulmonary exacerbations are defined in Section 4.7.4 and follow-up time is computed as detailed in Section 4.1.7.

## 4.7.2 Normality Assumption Checking

Not applicable.

# 4.7.3 Closed Testing Procedure for Primary Analysis

Not applicable.

## 4.7.4 Method of Analysis for Primary Endpoint

The NCFB pulmonary exacerbations collected from the Pulmonary Exacerbation eCRF form will be considered for the analysis. All cases in which the variable "Do these symptoms meet the protocol-defined criteria for NCFB pulmonary exacerbation?" is not consistent with data collected in the corresponding eCRF Pulmonary Exacerbations Symptoms form will be

| Sponsor: Zambon S.p.A. | Protocol Number: | Z7224L02 |
|------------------------|------------------|----------|
|------------------------|------------------|----------|

discussed during the blind review meeting. The decisions taken will be documented in the Blind Data Review and Analysis Sets Report.

The start of a protocol-defined NCFB pulmonary exacerbation will be taken as the first day that at least 3 of the 8 defining symptoms occurred concurrently for at least 24 hours as determined by the Investigator, as documented by the start date of the corresponding AE in the eCRF Adverse Events form and reviewed, where necessary, by the DAC (see Section 4.2.1) taking into consideration aspects such as start/stop date and associated systemic antibiotic therapy/hospitalisations.

Only NCFB pulmonary exacerbations with start date  $\geq$  date of first IMP dose and  $\leq$  date of treatment completion/discontinuation will be considered in the analysis. NCFB pulmonary exacerbations with start date = date of first IMP dose will be discussed on a case-by-case basis during the blind review of the data in order to evaluate whether they should be classified as having occurred in the screening period. The decisions taken will be documented in the Blind Data Review and Analysis Sets Report.

Resolution of a NCFB pulmonary exacerbation is defined as the date of completion of the required course(s) of antibiotic treatment, as collected in the eCRF Systemic Antibiotic Therapy form, and/or the Investigator's judgement that the NCFB pulmonary exacerbation has resolved, as documented by the end date provided for the corresponding AE in the eCRF Adverse Events form, whichever is the later of the two dates. If more than one systemic antibiotic therapy is administered for a NCFB pulmonary exacerbation, then the latest end date will be considered as the date of completion of the required course of antibiotic treatment.

In the case of a partial onset date of NCFB pulmonary exacerbation due to missing day, the onset of the event will be assumed to be the first day of the month. If the resultant derived date is prior to the date of first IMP dose, then it will be assumed to be equal to the first IMP dose date. Resultant derived dates will be reviewed during the blind review meeting and documented in the Blind Data Review and Analysis Sets Report.

In case of a partial resolution date of NCFB pulmonary exacerbation due to missing day, the resolution of the event will be assumed to be the last day of the month. If the resultant derived date is after the treatment completion/discontinuation date, then it will be assumed to be equal to the treatment completion/discontinuation date.

In case a NCFB pulmonary exacerbation presents a symptom with missing duration, following a conservative approach, the longest duration based on the start and stop dates of that symptom and until the resolution date of the NCFB pulmonary exacerbation will be imputed.

Two NCFB pulmonary exacerbations will be considered as a single episode in the statistical analysis if the second exacerbation started less than 14 days after the end of the systemic antibiotic therapy for the previous exacerbation (start date of the exacerbation - end date of the treatment of the previous exacerbation < 14 days). In case of more than two exacerbations for the same subject, this rule will be applied iteratively (therefore, more than two exacerbations may be considered as a single episode). Such cases will be discussed during the blind review of the data and the decisions taken will be documented in the Blind Data Review and Analysis Sets Report.

The above rule will not apply to the analysis of NCFB pulmonary exacerbations as AEs in the safety analysis.

In case of NCFB pulmonary exacerbations considered as a single episode:

Sponsor: Zambon S.p.A. Protocol Number: Z7224L02

- the start date of the first event will be considered as the start date;
- the stop date of the last event will be considered as the stop date;
- a worst case approach will be considered for duration of symptoms and requirement of
  hospitalisation. For example, if one of two exacerbations considered as a single episode
  has/have increased dyspnoea for ≥24 hours and <48 hours and the other one has
  increased dyspnoea for ≥ 48 hours, the single episode will be considered in the analysis
  as having dyspnoea for > 48 hours.

In order to investigate whether the use of inhaled colistimethate sodium reduces the frequency of pulmonary exacerbations compared to placebo in subjects with NCFB chronically infected with *P. aeruginosa*, the following hypothesis will be tested:

- Null hypothesis: there is no difference between inhaled colistimethate sodium and placebo as regards the effect on the pulmonary exacerbation rate
- Alternative hypothesis: inhaled colistimethate sodium reduces the pulmonary exacerbation rate in favour of inhaled colistimethate sodium compared to placebo.

The null hypothesis must be rejected for the efficacy of inhaled colistimethate sodium to be considered demonstrated.

The number and the percentage of subjects with NCFB pulmonary exacerbations, the number of NCFB pulmonary exacerbations and the total follow-up time in years, as defined in Section 4.1.7, will be summarised by treatment group.

The number of NCFB pulmonary exacerbations during the treatment period will be analysed using a negative binomial model including treatment, country, as detailed in Section 4.9.1, and use of stable concomitant therapy with oral macrolides as fixed effects and log-exposure time on treatment as an offset. The log-time on treatment in years will be calculated as ln (exposure time).

The adjusted mean annual NCFB pulmonary exacerbation rates in each treatment group and the adjusted rate ratio with their 95% CIs will be estimated by the model. OBSMARGINS option will be used for the estimates. The number of subjects considered in the model will be provided by treatment group.

The number and the percentage of subjects with 0, 1, 2 or >2 pulmonary exacerbations will be presented.

The number and the percentage of subjects with pulmonary exacerbations, the number of pulmonary exacerbations will also be presented by treatment group for severe (defined as those requiring intravenous antibiotics and/or hospitalisation) and not severe exacerbations.

A simple summary of the annualised pulmonary exacerbation rate will be calculated across subjects for each treatment as  $\{\sum_{i}^{n_{j}} \operatorname{exacerbation}_{i} / \sum_{i}^{n_{j}} \operatorname{exposure}_{i}\}$  where j denotes randomised treatment group,  $i=1\dots n_{j}$  denotes the number of subjects, exacerbation<sub>i</sub> and exposure<sub>i</sub> denote the number of exacerbations and exposure time for subject i.

The total duration of systemic antibiotic therapy, overall and by route, will be summarised by treatment group using descriptive statistics for continuous variables as well as distribution frequencies for the following categorisations:

1-7 days;

| Sponsor: Zambon S.p.A. Protocol Number: Z7224 | L02 |
|-----------------------------------------------|-----|
|-----------------------------------------------|-----|

- 8-15 days;
- 16-30 days;
- >30 days;
- Not Evaluable.

The total duration of systemic antibiotic therapy will be summarised overall and by category.

The duration of systemic antibiotic therapy will be evaluated considering the start and end date of the therapy associated with the pulmonary exacerbation. The duration of each course of systemic antibiotic therapy will be calculated using the following formula:

• Duration (days) = stop date – start date +1

For exacerbations treated with more than one systemic treatment, the duration will be calculated by summing the duration of the associated treatments. The overlapping days will be counted only once.

It is expected that all systemic antibiotic therapy will have completed (i.e. will have a stop date) at the end of the study when data are final, as all therapy stop dates are required to be known in order to derive the resolution date of pulmonary exacerbations per the definition described earlier in this section.

In order to calculate the duration of each course of systemic antibiotic therapy, the following rules will be applied for partial dates of start and stop date of systemic antibiotic therapies:

For the start date:

- if only the day is missing, the first day of the month will be assumed. If the resulting derived date is prior to the start date of the exacerbation, then start date of therapy will be assumed to be equal to the start date of the pulmonary exacerbation.
- if the day and the month are missing, then the date will not be imputed and the duration will be classified as "Not Evaluable".

For the stop date:

- if only the day is missing, the last day of the month will be assumed;
- if the day and the month are missing, then the date will not be imputed and the duration will be classified as "Not Evaluable".

Resultant dates will be discussed during the blind review meeting and documented in the Blind Data Review and Analysis Sets Report.

The above summary/analysis will be performed using the mITT Population and, where appropriate, the PP Population. Results for the PP Population will be considered as supportive.

# 4.7.4.1 CCI Analysis Using Alternative Definition of NCFB Pulmonary Exacerbation

A CCI analysis will be conducted using an alternative definition of NCFB pulmonary exacerbation for the mITT Population. The re-classification of pulmonary exacerbations will

| Sponsor: Zambon S.p.A. | Protocol Number: | Z7224L02 |
|------------------------|------------------|----------|
|------------------------|------------------|----------|

be done during the blind review meeting and documented in the Blind Data Review and Analysis Set Report.

In this **COL** analysis, a NCFB pulmonary exacerbation is defined as deterioration in three or more of the following key symptoms for at least 48 hours:



Subjects experiencing NCFB pulmonary exacerbations according to this alternative definition will be identified as those subjects having:

- An AE on the eCRF Adverse Events form with a MedDRA coded Preferred Term of "infective exacerbation of bronchiectasis" that is at least 48 hours in duration (i.e. stop date of AE − start date of AE + 1 ≥ 2);
- At least 3 of the above symptoms on the eCRF Pulmonary Exacerbation Symptoms form for the Pulmonary Exacerbation Number corresponding to that AE, where those symptoms all occur between the start and stop dates of the AE;
- At least 1 therapy on the eCRF Systemic Antibiotic Therapy form for the Pulmonary Exacerbation Number corresponding to that AE.

Analysis will be conducted following the same rules and methods as detailed above for the main definition of NCFB pulmonary exacerbations.

# 4.7.4.2 Column Analysis for Missing Data

In order to assess the potential impact of missing data on the results of the primary efficacy analysis, Copy Reference and Tipping Point column analyses using multiple imputation (MI) will be performed on all mITT subjects based on the approach proposed by Keene et al. [1]

Since Promis II was curtailed early, not all subjects are expected to have 365 days follow-up as intended in the original trial design. The expected duration of exposure for some subjects will therefore be shorter than 365 days. Therefore, and prior to unblinding, the expected duration of exposure in years,  $t_j$ , will be determined for each subject,  $n = 1 \dots j$ , individually using their randomisation date,  $r_j$ , and the date of study closure, d, where d = 28FEB2022 and  $t_j = \min([d - r_j + 1]/365.25, 365/365.25)$ . For all subjects with a realised follow-up duration,  $f_j$ , shorter than  $t_j$ , ie. with  $f_j < t_j$ , for example, due to early withdrawal or dropout
| Sponsor: Zambon S.p.A. Protocol Number: Z7224L02 | Sponsor: | Zambon S.p.A. | Protocol Number: | Z7224L02 |
|---|---|---|---|---|
|---|---|---|---|---|

at time  $f_j$  relative to randomisation, the number of pulmonary exacerbations in the missing period of follow-up,  $t_j - f_j$ , will be imputed.

The number of potentially missing exacerbations per subject will be imputed to include the following variables: treatment, country, as detailed in Section 4.9.1, and use of stable concomitant therapy with oral macrolides.

The imputation will be performed according to the following strategies:

- (1) Copy reference: imputation of missing data in both randomised treatment groups based on the data distribution of data observed in the placebo group. This analysis mimics the case where discontinued subjects who were randomised to colistimethate sodium are assumed to instaneously transition to placebo and lose any effect conferred by colistimethate sodium.
- (2) Tipping Point Analysis. For this analysis, discontinued subjects who were randomised to colistimethate sodium or placebo are initially imputed assuming the best case that data are missing at random and the treatment effect, CI and p-value are extracted. The analysis is subsequently repeated but now applying a small detrimental effect,  $\delta$ , in the imputation of colistimethate sodium subjects with missing data and, again, the treatment effect, CI and p-value are extracted. This analysis is then repeated with an increasing penalisation of colistimethate sodium treated subjects by addition of a detrimental effect,  $2\delta$ ,  $3\delta$ ,...,  $k\delta$  in order to find the 'Tipping Point' being that degree of penalisation that leads to loss of statistical significance on the primary endpoint analysis.

A total of 20 imputed datasets will be generated with each analysed using the same NB model as described for the primary analysis. Log event rate and log event rate ratio estimates and associated SEs arising from these 20 imputed datasets will then be combined via PROC MIANALYZE using Rubin's rules [2].

# 4.7.4.3 Subgroup Analyses

The primary endpoint will be explored in a number of subgroups as described in Section 4.1.5.

For each subgroup class separately, e.g. sex with classes Female and Male, the primary analysis negative binomial model will be reapplied to the primary endpoint data but now with two additional terms included, one for the subgroup, e.g. sex, and one for the interaction between the subgroup and randomised treatment. From this model, the p-value for the subgroup by randomised treatment interaction will be extracted along with estimates of the exacerbation rate ratio, colistimethate sodium:placebo, for each subgroup class, e.g. the exacerbation rate ratio, colistimethate sodium:placebo, for females and for males. The CI and p-value for these estimated exacerbation rate ratios will also be extracted and presented.

The results from all subgroups analyses will be presented in a single Forest Plot. This plot will display the treatment effect for each level of each subgroup with the associated confidence intervals and the treatment interaction p-value.

| Sponsor: Zambon S.p.A. Protocol Number: Z7224 | L02 |
|-----------------------------------------------|-----|
|-----------------------------------------------|-----|

# 4.7.5 Secondary Endpoint Analysis

If the primary endpoint shows statistical significance, a hierarchical testing procedure will be applied to the secondary endpoints to provide control of the overall Type I Error. This order shall be:



No test will be considered significant in this hierarchy unless every earlier test in it, including that for the primary outcome, is significant.

For the purposes of this SAP, it is anticipated that only the time to first pulmonary exacerbation and CCI total scores will be analysed for the PP Population in addition to the mITT Population.

# 4.7.6 Methods of Analysis for Secondary Endpoints



pulmonary exacerbation - date of randomisation. (It should be noted that this differs slightly from the CCI

CCI

For time-to-event endpoints, generally the + 1 is not included because this overestimates the time by 1 day for every event.)

Subjects completing the trial without CCI or who are discontinued prematurely CCI will be considered as censored at the time of their last follow-up, i.e. at the date of treatment completion/discontinuation. For the analysis, the following formula will be applied:

• Censoring time (days) = (date of treatment completion/discontinuation - date randomisation)

The number of subjects with a first **CC** events will be summarised.

| Sponsor: | Zambon S.p.A. | Protocol Number: | Z7224L02 |
|---|---|---|---|
| A Cox proportional hazard regression model will be applied to the data to provide an estimate of the hazard ratio (HR), colistimethate sodium:placebo. The model will include treatment group, country, as detailed in Section 4.9.1, and use of stable concomitant therapy with oral macrolides as covariates. The HR and its associated 95% CI and p-value will be extracted from the model and presented. A supportive analysis will be conducted using the log-rank test and the associated p-value will be presented. | | | |
| The number of cumulative nu and the estima 95% CIs will | Kaplan-Meier estimates in each treatment group will be presented: median time to CI, 25 <sup>th</sup> and 75 <sup>th</sup> percentiles and the corresponding CIs will be tabulated. The number of CI ——————————————————————————————————— | | |
| The estimate Kaplan-Meier | | each group will be d | isplayed graphically using a |
| In order to provide the best estimates of the median time to first exacerbation, a Weibull accelerated failure time model will be applied to the data using CCI. The same terms as fitted in the Cox regression analysis will be fitted in the Weibull analysis. From the Weibull analysis, estimates of the median time to first exacerbation plus 95% CI will be extracted for each randomised treatment arm along with the ratio of median times and its 95% CI and p-value. | | | |
| The CCI endpoint will also be analysed in terms of subgroup 7, as explained in Section 4.1.5. | | | |
| CCI And | ulysis for the Effect of Conco | mitant Antibiotic Ther | rapy |
| to the Cox prowill be conducted. The list of n | portional hazard regression lected to determine if the use has any impact of medications coded to WHO antibiotics are included in Apple 1, the response of the properties of t | model so that the hazes of antibiotics for on the CO DDD Preferred Term ppendix 3. If any medit ponse to the question ?" on the CO | ns for antibiotics and anti-<br>cation in the list has a related |
| "No", the med included as a than a CCI | ication was not taken for a antibiotics used for condi | in the opinion of Cl tions other than a ling list that do not | the Investigator. If answered and will be |

| Sponsor: | Zambon S.p.A. | Protocol Number: | Z7224L02 |
|---|---|---|---|
| other to covaria • Support antibiotomic and the covariant of the covarian | han a <mark>CCI</mark><br>te.<br>tive Cox proportional haz | ards analysis with us<br>than a protocol-defin | any antibiotics for conditions<br>(Yes/No) as an additional<br>se of any anti-pseudomonal<br>and pulmonary exacerbation |
| 4.7.6.2 | CI | | |
| For the CCI | the following weights will | be calculated: | |
| • CCI | | | |
| Each domain s | core will be calculated as fo | llows: | |
| • CCI | | | |
| The total score | will be calculated as follow | rs: | |
| • CCI | | | |
| Missing data | will be dealt with as des | cribed in CCI | |
| Weights of eac | h item and other details for o | calculation are reported | d in <mark>CC</mark> |
| statistics inclu<br>7/EOT will be<br>reported. Due<br>schedule, not a<br>collected will blocks random | End of Treatment) will be ding 25 <sup>th</sup> and 75 <sup>th</sup> percentil presented separately. Resu to CTP amendments and ll the subjects have undergo be summarised jointly. Con isation list no imbalance bet | les. Visit 7 for complets for absolute change to the corresponding the same sequence asidering the presence of tween treatments is expected. | assessed at nent group using descriptive leted subjects only and Visit es from baseline will also be g changes in the procedures of assessments. All the values of a stratified and permutated pected. Visit 5, Visit 6 and Visit 7 |
| Change nom | ouseine in col | 10 at visit 3, visit 4, | visit 5, visit 6 and visit / |

(completed subjects only) and Visit 7/EOT will be analysed using a linear mixed model for repeated measures including treatment, visit, treatment-by-visit interaction, use of stable concomitant therapy with oral macrolides and country, as detailed in Section 4.9.1, as fixed effects and baseline value as covariate. An unstructured covariance matrix will be assumed and the Kenward-Roger adjustment will be used for the degrees of freedom. The least square means in each treatment group, the least square mean differences between treatments, their 95% CIs

and associated p-values overall and at each visit will be estimated by the model. The OBSMARGINS option will be used.

The above summaries/analyses will be performed using the mITT and PP Populations. Results for the PP Population will be considered as supportive.

#### Notes:

• While for Visit 2, Visit 4, Visit 5, Visit 6 and Visit 7 the 3-month version of the cell is used, for Visit 3, data are collected for the 4-week version. Visit 2 scores will not be included in the linear mixed model analysis but they will be included in the descriptive analysis.

Summary statistics of the CCI and absolute change from baseline will be provided by treatment group for each trial visit.

Due to CTP amendments and to the corresponding changes in the procedures schedule and due to differences in the schedule of assessments in the local versions of the CTP, not all the subjects have undergone the same sequence of laboratory assessments. All the values collected will be summarised jointly. Considering the presence of a stratified and permutated blocks randomisation list no imbalance between treatments is expected.

The CCI as determined by the CCI (Visit 2) to Day 28 (Visit 3) and Visit 7 for completed subjects only and Visit 7/EOT will be compared between the treatment groups by a linear mixed model for repeated measures including treatment, country, as detailed in Section 4.9.1, and use of stable concomitant therapy with oral macrolides as fixed effects and baseline value as covariate. Least square means in each treatment group, least square mean difference between treatments, their 95% CIs and associated p-value will be estimated. OBSMARGINS option will be used for least square means estimates.

The analysis of covariance model will include only complete cases. Column analysis might be added during the blind review meeting.

The above summaries/analyses will be performed using the mITT Population.



| Sponsor: | Zambon S.p.A. | Protocol Number: | Z7224L02 |
|---|---|---|---|
| | rate estimates will be extrac<br>atio and its 95% CI and p-va | | group from the model along |
| The above summary/analysis will be performed using the mITT Population. | | | |
| 4.7.6.5 | CCI | | |
| The time to fin for the CCI in Section 4.7 | | | nalysed in the same manner as<br>sing a log-rank test as detailed |
| The above sur | nmary/analysis will be perfo | ormed using the mITT | Population. |
| 4.7.6.6 | CCI | | |
| The CCI | | will be present | ted by treatment group. |
| The endpoint | quantity for each subject wil | ll be computed with the | e following formula: |
| of durat | ions of <mark>CC</mark> | • | (follow-up time [days] – sum ollow-up time [days] } . |
| Follow-up tim | ne will be computed as detail | led in Section 4.1.7. | |
| completion/di | scontinuation, i.e. out of the | er of days of du | date after the treatment<br>ration after the treatment<br>Il be subtracted from the sum |
| groups using and use of station each treatment | an ANCOVA model included<br>to ble concomitant therapy with<br>tent group, least square mean<br>value will be estimated. OF | ing treatment, country<br>oral macrolides as fixe<br>n difference between t | pared between the treatment, as detailed in Section 4.9.1, ed effects. Least square means reatments, their 95% CIs and will be used for least square |
| In addition, a | summary statistics table wil | l be produced to displa | y: |
| • For ea | ch treatment group: | | |
| 0 | The number of subjects w, and their: | ith at least one protoc | ol-defined CCI |
| | <ul> <li>Mean exposure time</li> </ul> | e (months); | |
| | <ul> <li>Total number of CC</li> </ul> | | ; |
| | <ul> <li>Mean number of the contract of th</li></ul> | I | |
| | <ul> <li>Mean duration of </li> </ul> | CI ; | |
| | <ul> <li>Total months CCI</li> </ul> | | |
| 0 | The number of subjects s, and their: | with zero protocol | -defined CCI |
| | <ul> <li>Mean exposure time</li> </ul> | e (months); | |
| | ■ Total months CCI | | |
| | | CONFIDENTIAL | |

| Sponsor: | Zambon S.p.A. | Protocol Number: | Z7224L02 |
|---|---|---|---|
| 0 | Overall total months [CC] | ; | |
| О | Mean time CCI | (months). | |
| • Differe | nce in mean time | between | n treatment groups; |
| • Ratio o | f mean time CCI | between trea | tment groups. |
| 4.7.6.7 | Cl | | |
| Total number | | CCI | |
| Total number | described overall and by tre | atment group.<br>patient will be compu | ated by summing CO |
| Total number | _ | | form. Number of CC |
| . Na | mely: | vill be computed consi | dering CCI |
| • CCI | | | |
| | | | _ |
| Where: | | | |
| • CCI | | = sum {[CC <br>.] / CC | |
| | | | t1) [(Date of Assessment i) –<br>Assessment i+1) – (Date of |
| | Coeff i = 1 if Employment s<br>ssment i, Coeff i = 0 otherw | | ed or Temporarily Employed |
| Satterthwaite | method <sup>[6]</sup> . The correspond | ling two-sided p-valu | oups t-test by means of the<br>e will be presented. Mean<br>cresponding 95% CI will also |
| The above sun | nmaries/analyses will be per | formed using the mIT | Γ Population. |
| Notes: | | | |
| | | | e only the subsequent period<br>(referred to in the formula as |
| - | otion that no change in the omputed for each assessment | | relies on the curs during the |
| 4.7.6.8 | CI | | |
| | vill be provided overall and<br>mber of subjects with at leas | | ercentages will be computed erbation. |

Sponsor: Zambon S.p.A. Protocol Number: Z7224L02 The total number of **CCI** per subject will be analysed using a negative binomial regression model in a similar manner as the primary endpoint with the exception that the (log) duration of subject follow up rather than the duration of exposure will be included as the offset variable. The annualised **CC** will be extracted from this model for both randomised treatment groups as well the ratio of CC , together with its associated 95% confidence interval and p-value. A summary table will present the number and percentages of subjects with at least [60] having: The total duration of CC ■ will be summarised by treatment group using descriptive statistics for continuous variables. This summary shall include a presentation for the following categorisations: cci days; cci days; cci days; Not Evaluable. In case of CCI , the duration of CC will be calculated using the following formula: Duration of CCI In case of missing CC will be or CCI the CCI classified as "Not Evaluable". The above summaries/analyses will be performed using the mITT Population. 4.7.6.9 CCI For the column, the score for the following domains will be calculated as follows: : items 1, 2, 3, 4, 16; : items 17, 20, 25, 27, 28; items 6, 8, 9; : items 7, 10, 11, 23; : items 18, 19, 22, 26; : items 12, 13, 14; : items 5, 15, 21, 24; : items 29, 30, 31, 32, 33, 34, 35, 36, 37. CONFIDENTIAL

| Sponsor: Zambon S.p.A. Protocol Number: Z7224 | L02 |
|-----------------------------------------------|-----|
|-----------------------------------------------|-----|

Details for calculations are reported in Appendix 2: CC Version 3.1.

The column domain scores assessed at Visits 3 - 7 (End of Treatment) will be summarised by treatment group using descriptive statistics including 25<sup>th</sup> and 75<sup>th</sup> percentiles. Results for absolute changes from baseline will also be reported. Due to CTP amendments and to the corresponding changes in the procedures schedule, not all the subjects have undergone the same sequence of assessments. All the values collected will be summarised jointly. Considering the presence of a stratified and permutated blocks randomisation list no imbalance between treatments is expected.

Change from baseline in each common domain score will be analysed using a linear mixed model for repeated measures including treatment, visit, treatment-by-visit interaction, use of stable concomitant therapy with oral macrolides and country, as detailed in common as fixed effects and baseline value as covariate. An unstructured covariance matrix will be assumed and the Kenward-Roger adjustment will be used for the degrees of freedom. The least square means in each treatment group, the least square mean differences between treatments, their 95% CIs and associated p-values overall and at each visit will be estimated by the model. The OBSMARGINS option will be used.

The above summaries/analyses will be performed using the mITT Population.

# 4.8 Safety Analysis

All safety variables will be summarised overall and by treatment group using the Safety Population.

The safety variables are:

- AEs;
- Spirometry results;
- CCI CCI
- Vital signs;
- Physical examination results;
- Haematology and clinical chemistry parameters;
- 12-lead ECG parameters.

#### 4.8.1 Adverse Events

An AE is "any untoward medical occurrence in a subject or clinical trial subject administered a medicinal product and which does not necessarily have a causal relationship with this treatment".

An AE will be regarded as treatment-emergent if it has an onset date on or after the date of first IMP dose. For AEs with onset date on day of first IMP dose, the variable "Prior to first IMP administration?" in the Adverse Events eCRF form will be considered. AEs prior to first IMP administration will be considered as non-treatment-emergent. All other AEs, i.e. AEs with negative or missing answers to the question "Prior to first IMP administration?" will be considered as TEAEs. Partially missing dates will be handled as outlined in Section 4.11. If an

| Sponsor: | Zambon S.p.A. | Protocol Number: | Z7224L02 |
|----------|---------------|------------------|----------|
|----------|---------------|------------------|----------|

AE has a partial or fully missing date, and it is unclear whether the AE is treatment-emergent, it will be assumed that it is.

Only TEAEs will be included in the AE and SAE summaries. Non-treatment-emergent events will be included in the subject listings and flagged but not included in the summaries.

A summary table will present the number and percentage of subjects reporting:

- Any TEAEs;
- Any TEAEs by severity;
- Any TEAEs by relationship to IMP;
- Any TEAEs by action taken with IMP;
- Any Serious TEAEs;
- Any Fatal TEAEs.

The number of events occurring will also be reported.

Related AEs are those events for which there is a reasonable possibility that the IMP caused the event. When relationship to IMP is missing for a TEAE it will be imputed to be drug-related. Every effort should be made to query the site for complete data entry prior to database lock.

Fatal AEs are those reported with an outcome of "Fatal".

The number (and percentage) of subjects experiencing at least one TEAE, along with the number of events occurring, will be summarised by MedDRA SOC and PT, overall and by maximum severity.

A subject with more than one occurrence of the same AE in a particular SOC or PT will be counted only once in the total of those experiencing AEs in that particular SOC or PT. Two AEs with the same SOC or PT will be considered as two different events when calculating the "number of events" in the tables.

For summaries by maximum severity, if a subject experiences more than one event in the same SOC and PT, the subject will be counted in the maximum severity but all the events will be reported in their severity level. Maximum severity will be ranked as follows: severe > moderate > mild > unknown.

#### 4.8.1.1 Subsets for AE Descriptive Presentation

- Separate summary tables by SOC and PT will be presented for treatment-emergent SAFs
- Separate summary tables by SOC and PT and by SOC, PT and maximum severity will be presented for related TEAEs.
- Separate summary tables by SOC and PT will be presented for treatment-emergent related SAEs.
- Separate summary tables by SOC and PT will be presented for treatment-emergent AEs
  leading to the permanent discontinuation of IMP. An AE leading to discontinuation is
  an AE with action taken with IMP equal to "Permanently discontinued".

| Sponsor: | Zambon S.p.A. | Protocol Number: | Z7224L02 |
|----------|---------------|------------------|----------|
|----------|---------------|------------------|----------|

- Separate summary tables by SOC and PT will be presented for treatment-emergent fatal SAEs.
- Treatment-emergent SAEs and fatal AEs will be listed separately.
- The most frequent MedDRA PTs (≥5% of subjects with events in any treatment group) will be presented overall and by treatment. PTs will be used for tabulation, sorted by decreasing overall frequency.

All other information collected will be listed, as appropriate. Additionally, listings will display relative day of AE onset.

The relative day of AE onset will be calculated as follows:

- For pre-treatment AEs:
  - o AE onset date date of first IMP dose (if AE onset date is completely known);
  - o missing (if AE onset date is incomplete or unknown).
- For TEAEs:
  - AE onset date date of first IMP dose +1 (if AE onset date is completely known);
  - o missing (if AE onset date is incomplete or unknown).

#### Notes:

- AEs will be coded using MedDRA version 19.1 or higher (please refer to the final Data Management Plan for the latest coding information).
- Terms will be displayed in descending overall frequency (and then alphabetically) of SOCs and in descending overall frequency (and then alphabetically) of PTs within each SOC.

# 4.8.2 Spirometry Results

The following spirometry parameters will be summarised for each visit, as applicable, by treatment group and overall:

- FEV<sub>1</sub> (L);
- Predicted FEV<sub>1</sub> (%);
- FVC (L);
- Predicted FVC (%);
- Change in FEV<sub>1</sub> (L) from pre-salbutamol/albuterol intake to 30 minutes post-IMP.

Absolute value and change from baseline at each visit will be described by means of summary statistics for continuous variables.

The number and percentages (along with exact 95% CIs) of subjects experiencing bronchospasm at Visit 7 (End of Treatment) following IMP administration as clinically (as collected in the Spirometry eCRF forms) or spirometrically (>15% decrease in FEV<sub>1</sub> from pre-

| Sponsor: Z | Zambon S.p.A. | Protocol Number: | Z7224L02 |
|------------|---------------|------------------|----------|
|------------|---------------|------------------|----------|

salbutamol/albuterol intake to 30 minutes post-IMP) determined will be summarised by treatment. The number of subjects experiencing bronchospasm at all other visits will be listed. The subject will be considered spirometrically to have had a bronchospasm if presenting >15% decrease in FEV<sub>1</sub> from pre-salbutamol/albuterol intake to 30 minutes post-IMP or a positive answer to the above question.

The relative risk for colistimethate sodium/placebo will be provided with 95% asymptotic CIs. Treatment differences will be assessed using a Fisher Exact test. Subjects with no available result will be excluded from the analysis.

#### Notes:

- Change in FEV<sub>1</sub> (L) will be calculated as FEV<sub>1</sub> 30 minutes post-IMP FEV<sub>1</sub> presalbutamol/albuterol intake;
- Percentage change in FEV<sub>1</sub> (%) will be calculated as 100\*(change in FEV<sub>1</sub> [L] / FEV<sub>1</sub> pre-salbutamol/albuterol intake).



The summary will be repeated by status of previous usage of colistimethate sodium/colistin as detailed in Section 4.1.5.

Missing data will not be imputed. A separate summary will be presented summarising the last available results for each subject.

## Notes:

- Based on data collected on the Non-CF Bronchiectasis History eCRF form regarding previous usage of colistimethate sodium/colistin, subjects will be classified into:
  - Without any previous usage of colistimethate sodium/colistin;
  - With previous usage of colistimethate sodium/colistin;
  - o With missing data regarding previous usage of colistimethate sodium/colistin.

# 4.8.4 Haematology, Clinical Chemistry and Renal Function Parameters

The following haematology and clinical chemistry (including renal function) parameters will be summarised.

| Category | Parameter | Unit |
|-------------|-------------|------|
| Haematology | Haemoglobin | g/L |
| | Haematocrit | L/L |

| Red Cell Count x10E12/L White Cell Count x10E9/L Neutrophils % Total Lymphocytes % Monocytes % Eosinophils % Basophils % Neutrophils (Abs) x10E9/L Total Lymphs (Abs) x10E9/L Total Lymphs (Abs) x10E9/L Eosinophils (Abs) x10E9/L Basophils (Abs) x10E9/L Eosinophils (Abs) x10E9/L Basophils (Abs) x10E9/L Basophils (Abs) x10E9/L Chemistry Sodium mmol/L Potassium mmol/L Chloride mmol/L Uric Acid mmol/L Bilirubin (Total) umol/L Bilirubin (Conj) umol/L AST U/L ALT U/L GGT U/L ALP (Alk Phos) U/L Calcium mmol/L Calcium mmol/L Amylase U/L Renal Function BUN (Urea) mmol/L | Sponsor: | Zambon S.p.A. | Protocol Number: | Z7224L02 |
|---|---|---|---|---|
| White Cell Count Neutrophils % Total Lymphocytes % Monocytes % Eosinophils % Basophils % Neutrophils (Abs) x10E9/L Total Lymphs (Abs) x10E9/L Total Lymphs (Abs) x10E9/L Eosinophils (Abs) x10E9/L Eosinophils (Abs) x10E9/L Eosinophils (Abs) x10E9/L Basophils (Abs) x10E9/L Basophils (Abs) x10E9/L Chemistry Sodium mmol/L Potassium mmol/L Chloride mmol/L Uric Acid mmol/L Bilirubin (Total) mmol/L Bilirubin (Conj) mmol/L AST U/L ALT U/L GGT U/L ALP (Alk Phos) U/L Calcium mmol/L Calcium mmol/L Calcium mmol/L Calcium mmol/L Calcium mmol/L Calcium mmol/L | | D 10 110 | 10510/5 | |
| Neutrophils % Total Lymphocytes % Monocytes % Eosinophils % Basophils % Neutrophils (Abs) x10E9/L Total Lymphs (Abs) x10E9/L Eosinophils (Abs) x10E9/L Eosinophils (Abs) x10E9/L Eosinophils (Abs) x10E9/L Basophils (Abs) x10E9/L Platelets x10E9/L Platelets x10E9/L Chemistry Sodium mmol/L Potassium mmol/L Chloride mmol/L Uric Acid mmol/L Bilirubin (Total) umol/L Bilirubin (Conj) umol/L AST U/L ALT U/L ALT U/L GGT U/L ALP (Alk Phos) U/L Calcium mmol/L Amylase U/L | | | | |
| Total Lymphocytes % Monocytes % Eosinophils % Basophils % Neutrophils (Abs) x10E9/L Total Lymphs (Abs) x10E9/L Eosinophils (Abs) x10E9/L Eosinophils (Abs) x10E9/L Basophils (Abs) x10E9/L Basophils (Abs) x10E9/L Platelets x10E9/L Platelets x10E9/L Chemistry Sodium mmol/L Potassium mmol/L Chloride mmol/L Uric Acid mmol/L Bilirubin (Total) umol/L Bilirubin (Conj) umol/L AST U/L ALT U/L ALT U/L GGT U/L ALP (Alk Phos) U/L Calcium mmol/L Amylase U//L | | | | |
| Monocytes % Eosinophils % Basophils % Neutrophils (Abs) x10E9/L Total Lymphs (Abs) x10E9/L (Abs) x10E9/L Eosinophils (Abs) x10E9/L Basophils (Abs) x10E9/L Basophils (Abs) x10E9/L Platelets x10E9/L Platelets x10E9/L Chemistry Sodium mmol/L Potassium mmol/L Chloride mmol/L Uric Acid mmol/L Bilirubin (Total) umol/L Bilirubin (Conj) umol/L AST U/L ALT U/L ALT U/L GGT U/L ALP (Alk Phos) U/L Calcium mmol/L Amylase U//L | | | | |
| Eosinophils % Basophils % Neutrophils (Abs) x10E9/L Total Lymphs (Abs) x10E9/L (Abs) x10E9/L Eosinophils (Abs) x10E9/L Eosinophils (Abs) x10E9/L Basophils (Abs) x10E9/L Platelets x10E9/L Platelets x10E9/L Othemistry Sodium mmol/L Potassium mmol/L Chloride mmol/L Uric Acid mmol/L Bilirubin (Total) umol/L Bilirubin (Conj) umol/L AST U/L ALT U/L GGT U/L ALP (Alk Phos) U/L Calcium mmol/L Amylase U/L | | | · - | |
| Basophils Neutrophils (Abs) x10E9/L | | | | |
| Neutrophils (Abs) x10E9/L Total Lymphs x10E9/L (Abs) x10E9/L Eosinophils (Abs) x10E9/L Eosinophils (Abs) x10E9/L Basophils (Abs) x10E9/L Platelets x10E9/L Platelets x10E9/L Potassium mmol/L Potassium mmol/L Chloride mmol/L Uric Acid mmol/L Bilirubin (Total) umol/L Bilirubin (Conj) umol/L AST U/L ALT U/L GGT U/L ALP (Alk Phos) U/L Calcium mmol/L Amylase U/L | | Eosinophils | <b>%</b> | |
| Total Lymphs (Abs) Monocytes (Abs) Eosinophils (Abs) Rasophils (Abs) Platelets x10E9/L Basophils (Abs) x10E9/L Platelets x10E9/L Platelets x10E9/L Chemistry Sodium mmol/L Potassium mmol/L Chloride mmol/L Uric Acid Bilirubin (Total) Bilirubin (Conj) mmol/L AST U/L ALT GGT U/L ALP (Alk Phos) U/L Calcium mmol/L Amylase U/L | | Basophils | % | |
| (Abs) X10E9/L Monocytes (Abs) X10E9/L Eosinophils (Abs) X10E9/L Basophils (Abs) X10E9/L Platelets X10E9/L Platelets X10E9/L Chemistry Sodium mmol/L Potassium mmol/L Chloride mmol/L Uric Acid mmol/L Bilirubin (Total) umol/L Bilirubin (Conj) umol/L AST U/L ALT U/L GGT U/L ALP (Alk Phos) U/L Calcium mmol/L Amylase U/L | | Neutrophils (Abs) | x10E9/L | |
| Eosinophils (Abs) x10E9/L Basophils (Abs) x10E9/L Platelets x10E9/L Chemistry Sodium mmol/L Potassium mmol/L Chloride mmol/L Uric Acid mmol/L Bilirubin (Total) umol/L Bilirubin (Conj) umol/L AST U/L ALT U/L GGT U/L ALP (Alk Phos) U/L Calcium mmol/L Amylase U/L | | 2 1 | x10E9/L | |
| Basophils (Abs) x10E9/L Platelets x10E9/L Chemistry Sodium mmol/L Potassium mmol/L Chloride mmol/L Uric Acid mmol/L Bilirubin (Total) umol/L Bilirubin (Conj) umol/L AST U/L ALT U/L GGT U/L ALP (Alk Phos) U/L Calcium mmol/L Amylase U/L | | Monocytes (Abs) | x10E9/L | |
| Platelets x10E9/L Chemistry Sodium mmol/L Potassium mmol/L Chloride mmol/L Uric Acid mmol/L Bilirubin (Total) umol/L Bilirubin (Conj) umol/L AST U/L ALT U/L GGT U/L ALP (Alk Phos) U/L Calcium mmol/L Amylase U/L | | Eosinophils (Abs) | x10E9/L | |
| Chemistry Sodium mmol/L Potassium mmol/L Chloride mmol/L Uric Acid mmol/L Bilirubin (Total) umol/L Bilirubin (Conj) umol/L AST U/L ALT U/L GGT U/L ALP (Alk Phos) U/L Calcium mmol/L Amylase U/L | | Basophils (Abs) | x10E9/L | |
| Potassium mmol/L Chloride mmol/L Uric Acid mmol/L Bilirubin (Total) umol/L Bilirubin (Conj) umol/L AST U/L ALT U/L GGT U/L ALP (Alk Phos) U/L Calcium mmol/L Amylase U/L | | Platelets | x10E9/L | |
| Chloride mmol/L Uric Acid mmol/L Bilirubin (Total) umol/L Bilirubin (Conj) umol/L AST U/L ALT U/L GGT U/L ALP (Alk Phos) U/L Calcium mmol/L Amylase U/L | Chemistry | Sodium | mmol/L | |
| Uric Acid mmol/L Bilirubin (Total) umol/L Bilirubin (Conj) umol/L AST U/L ALT U/L GGT U/L ALP (Alk Phos) U/L Calcium mmol/L Amylase U/L | | Potassium | mmol/L | |
| Bilirubin (Total) umol/L Bilirubin (Conj) umol/L AST U/L ALT U/L GGT U/L ALP (Alk Phos) U/L Calcium mmol/L Amylase U/L | | Chloride | mmol/L | |
| Bilirubin (Conj) umol/L AST U/L ALT U/L GGT U/L ALP (Alk Phos) U/L Calcium mmol/L Amylase U/L | | Uric Acid | mmol/L | |
| AST U/L ALT U/L GGT U/L ALP (Alk Phos) U/L Calcium mmol/L Amylase U/L | | Bilirubin (Total) | umol/L | |
| ALT U/L GGT U/L ALP (Alk Phos) U/L Calcium mmol/L Amylase U/L | | Bilirubin (Conj) | umol/L | |
| GGT U/L ALP (Alk Phos) U/L Calcium mmol/L Amylase U/L | | AST | U/L | |
| ALP (Alk Phos) U/L Calcium mmol/L Amylase U/L | | ALT | U/L | |
| Calcium mmol/L Amylase U/L | | GGT | U/L | |
| Amylase U/L | | ALP (Alk Phos) | U/L | |
| · | | Calcium | mmol/L | |
| Renal Function BUN (Urea) mmol/L | | Amylase | U/L | |
| | Renal Functio | n BUN (Urea) | mmol/L | |
| Creatinine umol/L | | Creatinine | umol/L | |

Results as assessed at each applicable visit will be summarised by treatment group and overall using descriptive statistics for continuous variables. Absolute and percentage changes from baseline will also be presented.

A shift table will also be provided presenting results as lower than, within and higher than the central laboratory normal range. This will show the shift from baseline to each post-baseline visit, as well as to the most extreme value (defined as the value furthest outside [below or above] the central laboratory normal range) at any visit after baseline, including unscheduled visits.

# Notes:

- Change from baseline for each parameter will be computed using the formula:
  - Change (unit) = (AVAL [unit] baseline AVAL [unit]);
- All results outside the central laboratory normal range will be flagged in the data listings;

| Sponsor: Zambon S.p.A. Protocol Number: Z7224L02 | Sponsor: | Zambon S.p.A. | Protocol Number: | Z7224L02 |
|---|---|---|---|---|
|---|---|---|---|---|

- Repeat laboratory results within a visit will replace the original value;
- Due to CTP amendments and to the corresponding changes in the procedures schedule
  and due to differences in the schedule of assessments in the local versions of the CTP,
  not all the subjects have undergone the same sequence of laboratory assessments. All
  the values collected will be summarised jointly. Considering the presence of a stratified
  and permutated blocks randomisation list, no imbalance between treatments is
  expected.

## 4.8.5 Vital Signs

Respiratory rate (breaths per minute), heart rate (beats per minute), systolic and diastolic blood pressure (mmHg) and body temperature (°C) will be summarised overall and by treatment group at each applicable visit by means of descriptive statistics. Absolute and percentage changes from baseline to each visit after the first IMP dose will also be summarised. The number and percentage of subjects with Normal, Abnormal NCS and Abnormal CS results will be presented.

A shift table will also be provided for the clinical assessment. This will show the shift from baseline to each post-baseline visit, as well as to the worst overall result assessed at any visit after baseline, including unscheduled visits.

Additionally, for the Visit 7 summary, statistics for weight (kg) and BMI (kg/m²) will be presented.

#### Notes:

- BMI will be computed as weight at Visit 7 (kg) / (height at Visit 1 [m<sup>2</sup>]);
- Change from baseline for each parameter will be computed using the formula:

Change (unit) = AVAL (unit) - baseline AVAL (unit);

Due to CTP amendments and to the corresponding changes in the procedures schedule
and due to differences in the schedule of assessments in the local versions of the CTP,
not all the subjects have undergone the same sequence of vital sign assessments. All
the values collected will be summarised jointly. Considering the presence of a stratified
and permutated blocks randomisation, list no imbalance between treatments is
expected.

# 4.8.6 Physical Examination Results

Physical Examination findings collected at each visit will be described by treatment group and overall presenting the number and percentage of subjects with Normal, Abnormal NCS and Abnormal CS results for each body system as per the eCRF. Results for other body systems collected, but not specified in the eCRF will be listed only.

A shift table will also be provided. This will show the shift from baseline to each post-baseline visit, as well as to the worst overall result assessed at any visit after baseline, including unscheduled visits.

| Sponsor: Zambon S.p.A. | Protocol Number: | Z7224L02 |
|------------------------|------------------|----------|
|------------------------|------------------|----------|

#### Notes:

Due to CTP amendments and to the corresponding changes in the procedures schedule
and due to differences in the schedule of assessments in the local versions of the CTP,
not all the subjects have undergone the same sequence of physical examinations. All
the values collected will be summarised jointly. Considering the presence of a stratified
and permutated blocks randomisation list, no unbalance between treatments is
expected.

#### 4.8.7 12-Lead ECG

The 12-lead ECG overall interpretation at Visit 1 and Visit 7 will be described by treatment group and overall presenting the number and percentage of subjects with Normal, Abnormal NCS and Abnormal CS results. A shift table will also be provided showing the change from baseline to Visit 7, as well as to the worst overall result assessed at any visit after baseline, including unscheduled visits.

# 4.8.8 Pregnancy Test

Results from dipstick urine pregnancy tests for women of child-bearing potential will be listed only.

#### 4.8.9 Other Data

All other data collected in the eCRF will be listed only.

# 4.9 Adjustment for Covariates

The adjusted mean annual NCFB pulmonary exacerbation rate will be estimated by a negative binomial model including treatment, use of stable concomitant therapy with oral macrolides (e.g. azithromycin or erythromycin or clarithromycin: Yes/No) and country, as detailed in Section 4.9.1, as fixed effects and log-time on treatment as an offset. An exploratory model will also be fitted considering the number of CCI requiring oral/intravenous antibiotics in the last 12 months prior to study entry.

The Cox proportional hazard regression model for **CCI** will include use of stable concomitant therapy with oral macrolides (e.g. azithromycin or erythromycin or clarithromycin: Yes/No) and country, as covariates.

In the analysis of color total score and color domain scores, a linear mixed model for repeated measures will be applied. This will include treatment, visit, treatment-by-visit interaction, use of stable concomitant therapy with oral macrolides (e.g. azithromycin or erythromycin or clarithromycin: Yes/No) and country, as fixed effects and baseline value as covariate.

The **CCI** will be analysed by means of a linear mixed model for repeated measures including treatment, country, and use of stable concomitant therapy with oral macrolides (azithromycin or erythromycin or clarithromycin: Yes/No) as fixed effects and baseline value as covariate.

| Sponsor: Zambon S.p.A. | Protocol Number: | Z7224L02 |
|------------------------|------------------|----------|
|------------------------|------------------|----------|

#### 4.9.1 Country Effects

Sites are too numerous to be fitted in any model based analysis, therefore sites will be clustered under country with country included in modelling as a fixed effect. Given the similarity in geographic characteristics and concomitant treatments used (other than oral macrolides: i.e. bronchodilators, corticosteroids, etc) this approach is considered reasonable.

Smaller countries, with very few subjects, will be grouped into a single 'Other' country category. Based upon blinded trial data, the smaller countries to be grouped together the under 'Other' category are: Germany (N=3), Greece (N=3), Israel (N=4), Italy (N=1), New Zealand (N=6) and Portugal (N=2)...

Any change from this strategy will be discussed at the blind review meeting and documented in the Blind Data Review and Analysis Sets Report.

# 4.10 Protocol Deviations

# 4.10.1 Major Protocol Deviation Criteria

Exact definitions of major protocol deviations affecting safety and efficacy analyses will be discussed at the blind review meeting and documented in the Blind Data Review and Analysis Sets Report. The Protocol Deviation and Non-Compliance Management Plan documents the process for identifying protocol deviations that would potentially exclude subjects from the PP Population.

If major protocol deviations occur as outlined in the criteria below, then the data from complete individual subjects, individual visits or individual evaluations will be excluded from the population of analysis as indicated.

Exclusion of subjects or observations from the analyses will be decided jointly by the CRO and Sponsor's Study Team prior to unblinding of the randomisation code and database release.

The subjects or observations to be excluded, and the reasons for their exclusion, will be documented and approved by the above-mentioned persons prior to database release. The documentation will be filed together with the remaining trial documentation.

The number of subjects in each analysis population will be reported. Major protocol deviations excluding subjects from any particular population will be described, reporting the number of protocol violators for each criterion. All major protocol deviations will be listed and summarised for all screened subjects.

Major protocol deviations will be classified according to the following categories:

- Concomitant Medication / Administration of Prohibited Medication;
- Inclusion or Exclusion Criteria;
- Informed Consent / ICF not signed or signed late;
- Informed Consent / Other;
- Investigational Product / Incorrect IMP kit given to subject;
- Investigational Product / IMP Dosing;
- Investigational Product / IMP Storage;

- Investigational Product / Other;
- Met Withdrawal Criteria but was not Withdrawn;
- Patient Privacy (PP) / PP not signed;
- Patient Privacy / Other;
- Randomization / Mis-stratification;
- Randomization / Multiple Randomizations;
- Randomization / Other:
- Randomization / Randomized Not Treated;
- Randomization / Treated and Not Randomized;
- SAE not reported or reported late;
- Study Procedure / Missed procedure;
- Study Procedure / Other;
- Study Procedure / Site Staff Authorization, Delegation, Training;
- Study Procedure / Subject compliance;
- Study Procedure / Unmasking (not per protocol);
- Study Procedure / Visit Missing;
- Study Procedure / Washout;
- Visit Window.

These categories may be amended or other categories may be added, but any changes will be made prior to database lock and will be documented in the Blind Data Review and Analysis Sets Report.

#### 4.10.2 Protocol Deviations

Deviations from the protocol will be documented on an ongoing basis by the study monitors and clinical research associates or designee throughout the study period as detailed in the Protocol Deviation and Non-Compliance Management Plan.

At the time of database lock, prior to unblinding, the project manager or designee will forward all relevant documentation highlighting protocol deviations to the study statistician. These will be listed in the CTR. The study statistician will also verify occurrence of deviations from the protocol checking eCRF data, where feasible.

# 4.11 Missing Data

The validity of the negative binomial model planned for the primary efficacy analysis of the mean annual CCI relies on the MAR assumption. CCI have been outlined in Section 4.7.4.2 of this SAP to investigate the robustness of the primary endpoint conclusion under assumptions of MNAR.

| Sponsor: Zambon S.p.A. | Protocol Number: | Z7224L02 |
|------------------------|------------------|----------|
|------------------------|------------------|----------|

In the analysis of **CC** total score, **CC** domain scores and **CC** linear mixed models for repeated measures will be used to handle missing data. Under the MAR assumption, these models provide an unbiased estimate of the treatment effect that would have been observed if all subjects had continued on treatment [7].

analyses might be added during the blind review meeting if the amount of missing data makes it reasonable for further investigations of their influence on the overall study results. Decisions will be documented in the Blind Data Review and Analysis Sets Report.

Unless stated otherwise, there will be no imputation of missing values and only observed data will be included in the summaries.

The number of subjects with missing data will be presented under a "Missing" category. Unless otherwise stated, missing values will be included in the denominator count when computing percentages.

When continuous data are being summarised, only the non-missing values will be evaluated for computing summary statistics.

In order to calculate the duration of last usage of colistimethate sodium/colistin and the time from last administration of colistimethate sodium/colistin, the following rules will be applied for partial dates of start and stop date of last administration of colistimethate sodium/colistin:

For the start date:

- if only the day is missing, the first day of the month will be assumed;
- if the day and the month are missing, then the date will not be imputed and the time/duration will be classified as "Not Evaluable".

For the stop date:

- if only the day is missing, the last day of the month will be assumed;
- if the day and the month are missing, then the date will not be imputed and the time/duration will be classified as "Not Evaluable".

Where a medication start date is partially or fully missing, and it is unclear as to whether the medication is prior or concomitant, it will be assumed that it is concomitant.

In case of a partial onset date of a NCFB pulmonary exacerbation due to missing day, the onset of the event will be assumed as the first day of the month. If the resultant derived date is prior to the date of first IMP dose, then it will be assumed to be equal to the first IMP dose date.

In case of a partial resolution date of a NCFB pulmonary exacerbation due to missing day, the resolution of the event will be assumed as the last day of the month. If the resultant derived date is after the treatment completion/discontinuation date, then it will be assumed to be equal to the treatment completion/discontinuation date.

In case a NCFB pulmonary exacerbation presents a symptom with missing duration, following a conservative approach, the longest duration will be imputed.

In order to calculate the duration of each course of systemic antibiotic therapy, the following rules will be applied for partial dates of start and stop date of systemic antibiotic therapies:

For the start date:

| Sponsor: | Zambon S.p.A. | Protocol Number: | Z7224L02 |
|----------|---------------|------------------|----------|
|----------|---------------|------------------|----------|

- if only the day is missing, the first day of the month will be assumed. If the resulting derived date is prior to the start date of the exacerbation, then start date of therapy will be assumed to be equal to the start date of the exacerbation.
- if the day and the month are missing, then the date will not be imputed.

For the stop date:

- if only the day is missing, the last day of the month will be assumed.
- if the day and the month are missing, then the date will not be imputed and the duration will be classified as "Not Evaluable".

The domain scores of the considered non-missing if the following conditions are satisfied:

- Symptoms score: missing items ≤ 2;
- Activity score: missing items ≤ 4;
- Impacts score: missing items ≤ 6.

If at least one domain score is missing, the total score will be considered as missing.

The domain scores of **CC** will be considered non-missing if the responses are missing for half or less of the items in the domain.

If an AE has a partially or fully missing date, and it is unclear whether the AE is treatmentemergent, it will be assumed that it is. In the AEs analysis, when relationship to IMP is missing for a TEAE it will be imputed to be drug-related. Every effort should be made to query the site for complete data entry prior to database lock.

Other critical missing data, if any, will be discussed during the blind review of the data. Decisions will be fully documented in the Analysis Set Specifications Document.

# 4.12 Deviations from the SAP

Any deviations from the original SAP will be described and justified in the final CTR, whether written post interim or final analysis.

# 4.13 Changes in Conduct or Planned Analyses from the Protocol

Sections 2.2, 4.4.11, 4.7.5 and 4.7.6.3: The protocol incorrectly referred to the units for the determination of CCI which have been reported as CCI by the central laboratory.

Section 4.7.4: The protocol states that the Negative Binomial Model will consider the log-time on study as offset. However, as specified in Section 4.1.7, NCFB Pulmonary Exacerbations analyses focus on the treatment period so log-time on treatment will be considered.



| Sponsor: Zambon S.p.A. Protocol Number: Z7224L02 | Sponsor: | Zambon S.p.A. | Protocol Number: | Z7224L02 |
|---|---|---|---|---|
|---|---|---|---|---|

Section 4.7.6.1: The protocol states that the CCI

For time-

to-event endpoints, generally the + 1 is not included because this overestimates the time by 1 day for every event, therefore "+ 1" has been deleted.

Section 4.7.6.5: The protocol states that the column total score will be computed and analysed. However, as recommended in the Manual Scoring Instructions and the column domain scores will be presented and analysed.

There have been no other changes in analyses from those defined in the protocol.

# 4.14 Algorithms/SAS Codes

The SAS codes for descriptive statistics and frequency counts detailed below are examples only and other procedures may be used, if appropriate.

Tables that need descriptive statistics – continuous variables:

```
PROC UNIVARIATE DATA=dset NOPRINT;

VAR var1 var2 var3 ...varn;

BY byvar; (optional)

OUTPUT OUT= outset

N=n MEAN=mean MIN=min MAX=max MEDIAN=median STD=std *Q1=q1
Q3=q3; *Include Q1 and Q3 for CCT data only;
RUN;
```

Tables that need frequency counts:

```
PROC FREQ DATA=dset NOPRINT;
BY byvar; (optional)
TABLES var1*var2 /out= outset;
RUN:
```

Tables that need T-Test;

```
PROC TTEST DATA=dset;
CLASS var1;
VAR var1N;
RUN:
```

 Tables that need exact 95% CIs for risk difference between groups for proportions and Fisher's Exact:

```
PROC FREQ DATA=dset;
BY byvar; (optional)
TABLES var*treatment / MEASURES RISKDIFF EXACT ALPHA=0.05;
EXACT MEASURES;
OUTPUT OUT= outset EXACT MEASURES RISKDIFF;
WHERE wherever; (optional)
RUN;
```

• Tables that need 95% CIs within group for binomial proportions:

```
PROC FREQ DATA=dset;
BY byvar; (optional)
TABLES var1;
EXACT BINOMIAL;
OUTPUT OUT= outset BINOMIAL;
RUN;
```

• Tables that require analysis of (co)variance and 95% CIs between arms for continuous variables:

```
PROC GLM DATA= dset OUTSTAT=outset;
CLASS treatment psite med;
```

```
MODEL change = treatment psite med baseline/ SOLUTION;

LSMEANS treatment / STDERR PDIFF CL OBSMARGINS;

BY byvar; (optional)

WHERE wherever; (optional)

RUN;
```

# Notes:

- Psite represents the country, as detailed in Section 4.9.1;
- Med represents use of stable concomitant therapy with oral macrolides (e.g. azithromycin or erythromycin or clarithromycin) (Yes/No);
- Change represents the change from baseline of the variable;
- Baseline represents the baseline value of the variable;
- Treatment order: 1= Colistimethate Sodium, 2= Placebo.
- Tables that require Kaplan-Meier estimates and log-rank test:

```
PROC LIFETEST DATA=dset OUTSURV=LIFE METHOD=KM timelist=(0 28 90 180 270 EoT) reduceout;

TIME time*event (1);

ID subject;

STRATA treatment;

WHERE wherever; (optional)

RUN;
```

#### Notes:

- Time represents the time to event or time to censoring;
- Event represents the censoring indicator (1 = censored);
- EoT should be replaced by the last time (in days) to event >270 days (if any);

# Tables that require Cox proportional hazards model and 95% CIs of hazard ratios between treatments:

```
PROC PHREG data=dset;

CLASS treatment psite med;

MODEL time*event(1) = treatment psite med / ties=exact;

HAZARDRATIO 'Col. Sodium vs Placebo' treatment / cl=both;

BY byvar; (optional)

WHERE wherever; (optional)

RUN;
```

#### Notes:

- Psite represents the country, as detailed in Section 4.9.1;
- Med represents use of stable concomitant therapy with oral macrolides (e.g. azithromycin or erythromycin or clarithromycin) (Yes/No);
- Time represents the time to event or time to censoring:
- Event represents the censoring indicator (1 = censored);
- If the option ties=exact requires a considerable amount of computer resources, the Efron approximation will be used (ties=efron).
- Treatment order: 1= Colistimethate Sodium, 2= Placebo.

# Tables that require negative binomial modelling, including 95% CIs of treatment ratios:

```
PROC GENMOD data = dset;

CLASS treatment psite med;

MODEL count = treatment psite med / offset=log_years link=log dist=negbin wald type3;

ESTIMATE 'Col. Sodium / Placebo' treatment 1 -1 / exp;

Ismeans treatment / ilink cl diff exp om;

BY byvar; (optional)

WHERE wherever; (optional)

RUN;
```

#### Notes:

- Psite represents the country, as detailed in Section 4.9.1;
- Med represents use of stable concomitant therapy with oral macrolides (e.g. azithromycin or erythromycin or clarithromycin) (Yes/No);
- Count represents the total number of exacerbations for each patient;
- log years represents the logarithm of the follow-up time in years;
- Treatment order: 1= Colistimethate Sodium, 2= Placebo.
- Tables that require linear mixed model for repeated measures and 95% CIs of differences between treatments:

```
PROC\ MIXED\ data = dset;
   CLASS treatment visit psite med sub;
   MODEL change = treatment visit treatment*visit psite med baseline/ s ddfm=kr;
   REPEATED visit / subject=sub type=un r;
   LSMEANS treatment treatment*visit / om at means cl slice=visit;
   LSMESTIMATE treatment
       'Col. Sodium / Placebo'
                               1 - 1 / cl;
   LSMESTIMATE treatment*visit
       'Col. Sodium / Placebo: Visit 4' 1 0 0 0 -1 0 0 0,
       'Col. Sodium / Placebo: Visit 5' 0 1 0 0 0 -1 0 0.
       'Col. Sodium / Placebo: Visit 6' 0 0 1 0 0 0 -1 0,
       'Col. Sodium / Placebo: Visit 7' 0 0 0 1 0 0 0 -1/cl;
   BY byvar; (optional)
   WHERE wherever; (optional)
RUN;
```

# Notes:

- Visit represents the clinic visit;
- Psite represents the country, as detailed in Section 4.9.1;
- Med represents use of stable concomitant therapy with oral macrolides (e.g. azithromycin or erythromycin or clarithromycin) (Yes/No);
- Sub represents the Subject Number;
- Change represents the change from baseline to each visit of the variable;
- Baseline represents the baseline value of the variable;
- Treatment order: 1= Colistimethate Sodium, 2= Placebo.

\_

# • Multiple Imputation for pulmonary exacerbation rate

An example of SAS code is provided below for the CCI and analyses pulmonary exacerbation rate.

# Missing at random and copy reference imputation

ORDER BY Iteration, Subject;

```
PROC GENMOD DATA=dataset1act; /* Colistimethate Sodium subjects */
   MODEL count = treatment d psite_d1-psite_dx med_d / OFFSET=log_years
   DIST=NEGBIN;
   /* >1000 imputations since some will be discarded due to convergence issues with the
   model */
   BAYES NBI=1000 NMC=11000 THIN=10 OUTPOST=dataset2act SEED=34783129;
RUN;
DATA dataset3act;
   SET dataset2act;
   RENAME treatment d = c treatment d
            psite d1-psite dx=c psite d1-c psite dx
            med d=c med d;
RUN:
PROC GENMOD DATA=dataset1plb; /* Placebo subjects */
   MODEL count = treatment d psite d1-psite dx med d / OFFSET=log years
   DIST=NEGBIN;
   /* >1000 imputations since some will be discarded due to convergence issues with the
   model */
   BAYES NBI=1000 NMC=11000 THIN=10 OUTPOST=dataset2plb SEED=34783129;
RUN;
DATA dataset3plb;
   SET dataset2plb;
   RENAME treatment d = c treatment d
            psite d1-psite dx=c psite d1-c psite dx
            med d=c med d;
RUN;
PROC SQL;
   CREATE TABLE dataset4act mar AS
   SELECT dataset1act.*, dataset3act.*
   FROM dataset1act, dataset3act
   ORDER BY Iteration, Subject;
   CREATE TABLE dataset4act cr AS
   SELECT dataset1act.*, dataset3plb.*
   FROM dataset1act, dataset3plb
```

```
CREATE TABLE dataset4plb AS
    SELECT dataset1plb.*, dataset3plb.*
    FROM dataset1plb, dataset3plb
    ORDER BY Iteration, Subject;
QUIT;
DATA dataset4all mar; /* For Missing at Random */
   SET dataset4act mar dataset4plb;
   BY Iteration Subject;
RUN;
DATA dataset4all cr; /* For Copy Reference */
   SET dataset4act cr dataset4plb;
   BY Iteration Subject;
RUN:
DATA dataset5 mar; /* Missing at Random */
    SET dataset4all mar;
   BY Iteration Subject;
   ARRAY c[*] c psite d1-c psite dx c med d;
   ARRAY x[*] psite_d1-psite_dx med_d;
   k=1/Dispersion;
    imp\ subj = (vears < 365/365.25);
   years imp=MAX(years, years exp);
    log years imp=LOG(years imp);
    linpred 1=.;
   IF imp subj THEN DO;
      years miss=years imp-years;
      linpred_1=Intercept;
      DO i=1 TO DIM(c);
          linpred 1+c[i]*x[i];
      END:
      linpred mar=linpred 1+c treatment d*treatment d;
      v2hat mar=years miss*EXP(linpred mar);
      CALL STREAMINIT(3231212);
      y2 mar=RAND('NEGBINOMIAL',k/(k+y2hat mar),k);
      y_imp_mar=count+y2 mar;
   END;
    ELSE DO;
      y imp mar=count;
   END;
RUN:
DATA dataset5 cr; /* Copy Reference */
    SET dataset4all cr;
    BY Iteration Subject;
   ARRAY c[*] c psite d1-c psite dx c med d;
```

```
ARRAY x[*] psite d1-psite dx med d;
    k=1/Dispersion;
    imp subj=(years<365/365.25);
   years imp=MAX(years, years exp);
    log years imp=LOG(years imp);
    linpred 1=.;
   IF imp subj THEN DO;
      years miss=years imp-years;
      linpred 1=Intercept;
      DO i=1 TO DIM(c);
          linpred 1+c[i]*x[i];
      END:
      lingred cr=lingred 1+c treatment d;
      y2hat cr=years miss*EXP(linpred cr);
      CALL STREAMINIT(3231212);
      v2 cr = RAND('NEGBINOMIAL', k/(k+v2hat cr), k);
      v imp cr = count + v2 cr;
    END;
    ELSE DO;
      y imp cr=count;
    END:
RUN:
```

#### Notes:

- dataset1 includes one record per patient;
- treatment represents the treatment group (treatment order: 1 = colistimethate sodium, 2 = placebo);
- treatment\_d represent the dummy variables for treatment group (values of the dummy variables: 0 for colistimethate sodium; 1 for placebo);
- Psite represents the country, as detailed in Section 4.9.1;
- psite d1-psite dx represent the dummy variables for the country;
- Med represents use of stable concomitant therapy with oral macrolides (e.g. azithromycin or erythromycin or clarithromycin) (Yes/No);
- med\_d represents the dummy variable for use of stable concomitant therapy with oral macrolides;
- years represents the observed follow-up time in years;
- years exp represents the expected follow-up time in years
- log years represents the logarithm of the follow-up time in years.

#### Analysis step

The imputed dataset obtained using the above SAS code will be finally analysed and the results will be combined.

```
ODS OUTPUT LSMeans=lsmeans_mar Estimates=ratios_mar; /* Missing at Random */
PROC GENMOD DATA=dataset5_mar;
BY Iteration;
```

```
Sponsor:
             Zambon S.p.A.
                                      Protocol Number:
                                                         Z7224L02
    CLASS treatment psite med;
   /* MAR imputation */
   MODEL y imp mar = treatment psite med/OFFSET=log years imp DIST=NEGBIN;
   LSMEANS treatment / ilink cl diff exp om;
      ESTIMATE 'Col. Sodium / Placebo' treatment 1 -1 / exp;
RUN:
DATA lsmeans mar2;
    SET lsmeans mar (WHERE=(zValue ne .));
    BY Iteration;
   IF first.Iteration THEN Imputation +1;
   IF Imputation LE 1000;
RUN;
ODS OUTPUT ParameterEstimates=lsmeans mar3;
PROC MIANALYZE PARMS=lsmeans mar2;
    CLASS treatment;
   MODELEFFECTS treatment;
RUN;
DATA lsmeans mar4;
    SET lsmeans mar3;
    exp est=EXP(Estimate);
    exp lcl=EXP(LCLMean);
    exp ucl=EXP(UCLMean);
RUN;
DATA ratios mar2 (RENAME=LBetaEstimate=Estimate);
    SET ratios mar (WHERE=(ChiSq ne .));
   BY Iteration;
   IF first.Iteration THEN Imputation +1;
   IF Imputation LE 1000;
   Effect='Label';
RUN;
ODS OUTPUT ParameterEstimates=ratios mar3;
PROC\ MIANALYZE\ PARMS = ratios\ mar2;
    CLASS Label;
    MODELEFFECTS Label:
RUN;
DATA ratios mar4;
    SET ratios mar3;
    exp est=EXP(Estimate);
    exp\ lcl = EXP\ (LCLMean);
    exp\ ucl = EXP\ (UCLMean);
RUN:
```

```
ODS OUTPUT LSMeans=Ismeans cr Estimates=ratios cr; /* Copy Reference */
PROC GENMOD DATA=dataset5 cr;
    BY Iteration;
    CLASS treatment psite med;
   /* CR imputation */
   MODEL\ y\ imp\ cr = treatment\ psite\ med/\ OFFSET=log\ years\ imp\ DIST=NEGBIN;
   LSMEANS treatment / ilink cl diff exp om;
      ESTIMATE 'Col. Sodium / Placebo' treatment 1 -1 / exp;
RUN;
DATA lsmeans cr2;
    SET lsmeans cr (WHERE=(zValue ne .));
   BY Iteration;
   IF first.Iteration THEN Imputation +1;
   IF Imputation LE 1000;
RUN:
ODS OUTPUT ParameterEstimates=lsmeans cr3;
PROC MIANALYZE PARMS=lsmeans cr2;
    CLASS treatment;
   MODELEFFECTS treatment;
RUN;
DATA lsmeans cr4;
    SET Ismeans cr3;
    exp est=EXP(Estimate);
    exp lcl=EXP(LCLMean);
    exp ucl=EXP(UCLMean);
RUN:
DATA ratios cr2 (RENAME=LBetaEstimate=Estimate);
    SET ratios cr (WHERE=(ChiSq ne .));
   BY Iteration:
   IF first.Iteration THEN _Imputation_+1;
   IF Imputation LE 1000;
   Effect='Label';
RUN;
ODS OUTPUT ParameterEstimates=ratios cr3;
PROC MIANALYZE PARMS =ratios cr2;
    CLASS Label;
   MODELEFFECTS Label;
RUN:
DATA ratios cr4;
    SET ratios cr3;
    exp est=EXP(Estimate);
    exp\ lcl = EXP\ (LCLMean);
```

| Sponsor: | Zambon S.p.A. | Protocol Number: | Z7224L02 |
|----------|---------------|------------------|----------|

exp\_ucl= EXP (UCLMean);
RUN;

# 5 Tables and Listings

# 5.1 Table Format

All output will be produced using SAS version 9.4 or a later version.

- All TFLs will be produced in landscape format on American letter size, unless otherwise specified.
- All TFLs will be produced using the Courier New font, size 8, which is the smallest acceptable point size for the Regulatory Authorities.
- The data displays for all TFLs will have a minimum blank 1-inch margin on all 4 sides.
- Headers and footers for figures will be in Courier New font, size 8 which is the smallest acceptable point size for the Regulatory Authorities.
- Legends will be used for all figures with more than 1 variable, group, or item displayed.
- TFLs will be in black and white (no colour).
- Specialized text styles, such as bolding, italics, borders, shading, and superscripted and subscripted text, will not be used in the TFLs, unless otherwise specified. On some occasions, superscripts 1, 2, or 3 may be used (see below).
- Only standard keyboard characters will be used in the TFLs. Special characters, such as non-printable control characters, printer-specific, or font-specific characters, will not be used. Hexadecimal-derived characters will be used, where possible, if they are appropriate to help display math symbols (e.g., μ). Certain subscripts and superscripts (e.g., cm², C<sub>max</sub>) may be employed on a case-by-case basis.
- Mixed case will be used for all titles, footnotes, column headers, and programmersupplied formats, as appropriate.

#### Headers

• All output should have the following header at the top left of each page:

Zambon Protocol Z7224L02 (CCI

• All output should specify the Draft/Final Run status at the top centre of each page.

| Sponsor: | Zambon S.p.A. | Protocol Number: | Z7224L02 |
|----------|---------------|------------------|----------|
|----------|---------------|------------------|----------|

- All output should have Page n of N at the top right corner of each page. TFLs are
  internally paginated in relation to the total length (i.e., the page number should appear
  sequentially as page n of N, where N is the total number of pages in the table).
- The date output was generated should appear along with the program name as a footer on each page.

# **Display Titles**

• Each output is identified by the designation and a numeral. (i.e., Table 14.1.1). ICH E3 numbering is strongly recommended. A decimal system (x.y and x.y.z) is used to identify TFLs with related contents. All titles will be centre-aligned. The analysis population will be identified on the line immediately following the title. The output number and title will be single-line spaced. A solid line spanning the margins will separate the display titles from the column headers. There will be one blank line between the last title and the solid line.

# Table x.y.z First Line of Title Second Line of Title if Needed

(mITT Population)

In a listing, in the case that a subject's record has been continued to the next page, an appropriate identification (e.g., the subject ID number) must be presented at the beginning of that page.

# 5.2 Conventions

Unless otherwise specified, in summary tables of continuous variables, the minimum and maximum values will be displayed to the same number of decimal places as the raw data, the mean and median will be presented to one extra decimal place compared to the raw data, and the standard deviation will be displayed to two extra decimal places compared to the raw data. Wherever possible data will be decimal aligned.

Unless otherwise specified, frequency tabulations will be presented by number and percentage, where the percentage is presented in brackets to 1 decimal place. Percentages between 0.05% and 0.1% will be rounded to 0.1%. Percentages less than 0.05% will be displayed as <0.1%. Percentages between 99.90% and 99.95% will be rounded to 99.9%. Percentages more than 99.95% will be displayed as >99.9%.

P-values, if applicable, will be presented to 5 decimal places. If the p-value is less than 0.00001 then it will be presented as <0.00001. If the rounded result is a value of 1.00000, it will be displayed as >0.99999.

Any date information in the listing will use the *date9*. format, for example, 07MAY2002. In the listing, a unit associated with a variable will be presented only once within parentheses either below or next to that variable in the heading portion.

| Sponsor: Zambon S.p.A. | Protocol Number: | Z7224L02 |
|------------------------|------------------|----------|
|------------------------|------------------|----------|

Unless otherwise specified, listings should be sorted by treatment group, subject and visit and have the source ADaM dataset referenced in a footnote.

All tables, listings and figures will be converted into Rich text format with the format/file extension specified and collated into three separate complete documents. The combined documents will be in .pdf format.

| | Sponsor: | Zambon S.p.A. | Protocol Number: | Z7224L02 |
|-----|----------|---------------|------------------|----------|
| - 1 | | | | |

# 5.3 Tables

# 5.3.1 Section 14.1: Demographic and Baseline

# 5.3.2 Section 14.2: Primary

| Table 14.2.1.1.1.1 | NCFB Pulmonary Exacerbations: Mean Annual Rate by Negative Binomial Model | (mITT Population) |
|---|---|---|
| Table 14.2.1.1.1.2 | NCFB Pulmonary Exacerbations: Mean Annual Rate by Negative Binomial Model by Country | (mITT Population) |

| Sponsor: | Zambon S.p.A. | Protocol Number: | Z7224L02 | |
|---|---|---|---|---|
| Table 14.2.1.1.2 | NCFB Pulmonary Exacerbations: Mean Ann | • 0 | | (PP Population) |
| Table 14.2.1.1.3 | NCFB Pulmonary Exacerbations: Mean A Definition of Pulmonary Exacerbation | nnual Rate by Negative Binomial | Model - Alternative | (mITT Population) |
| Table 14.2.1.1.4.1 | NCFB Pulmonary Exacerbations: Mean Annu for Missing Data | nal Rate by Negative Binomial Model | - CCI Analysis | (mITT Population) |
| Table 14.2.1.1.4.2 | NCFB Pulmonary Exacerbations: Mean An<br>Analysis | mual Rate by Negative Binomial M | Iodel - Tipping Point | (mITT Population) |
| Table 14.2.1.1.5 | NCFB Pulmonary Exacerbations: Mean Ann | ual Rate by Negative Binomial Mode | l by IMP Adherence | (mITT Population) |
| Table 14.2.1.1.6 | NCFB Pulmonary Exacerbations: Mean A Pulmonary Exacerbations in the 12 Months F | | Model – Number of | (mITT Population) |
| Table 14.2.1.1.7 | NCFB Pulmonary Exacerbations: Mean Ar<br>Pulmonary Exacerbations Requiring Oral or<br>Entry | | | (mITT Population) |
| Table 14.2.1.1.8 | NCFB Pulmonary Exacerbations: Mean Annu<br>Colistimethate Sodium/Colistin | ual Rate by Negative Binomial Model | by Previous Usage of | (mITT Population) |
| Table 14.2.1.1.9 Table 14.2.1.1.10 Table 14.2.1.2.1 Table 14.2.1.2.2 Table 14.2.1.3 | NCFB Pulmonary Exacerbations: Mean Ann<br>NCFB Pulmonary Exacerbations: Mean Ann<br>NCFB Pulmonary Exacerbations: Unadjusted<br>NCFB Pulmonary Exacerbations: Systemic Annual Pulmonary Exacerbations: Systemic An | ual Rate by Negative Binomial Mode<br>I Mean Annual Rate Overall and by S<br>I Mean Annual Rate Overall and by S | l by Gender<br>Severity | (mITT Population)<br>(mITT Population)<br>(mITT Population)<br>(PP Population) |
| 14016 14.2.1.3 | NCFB Pulmonary Exacerbations: Systemic A | Midolotic Therapy | | (mITT Population) |

# 5.3.3 Section 14.2: Secondary

| Table 14.2.2.1.1 | CCI | : Kaplan-Meier Estimates | (mITT Population) |
|---|---|---|---|
| Table 14.2.2.1.2 | CCI | : Kaplan-Meier Estimates | (PP Population) |
| Table 14.2.2.1.5 | CCI | : Weibull Accelerated Failure Time Model | (mITT Population) |
| Table 14.2.2.1.6 | CCI | : Weibull Accelerated Failure Time Model | (PP Population) |
| Table 14.2.2.2.1 | CCI | : Cox proportional hazard regression model | (mITT Population) |
| Table 14.2.2.2.2 | CCI | : Cox proportional hazard regression model | (PP Population) |
| Table 14.2.2.2.3 | Analysis for the Effect of Concomitant A | : Cox proportional hazard regression model - CC | (mITT Population) |
| | Analysis for the Effect of Concomitant A | Aminonic incrapy | • |

| Sponsor: | Zambon S.p.A. | Protocol Number: | Z7224L02 | |
|---|---|---|---|---|
| Table 14.2.2.2.4 | CCI Analysis for the Effect of | : Cox proportional hazard re<br>Concomitant Anti-Pseudomonal Antibiotic The | | (mITT Population) |
| Table 14.2.2.3 | CCI | : Kaplan-Meier Estimates by | | (mITT Population) |
| Table 14.2.2.5.1 | : Domain Scores at | nd Total Score Results and Change Versus Base | | (mITT Population) |
| Table 14.2.2.5.2 | : Domain Scores at | nd Total Score Results and Change Versus Basel | line | (PP Population) |
| Table 14.2.2.5.3 | : Linear Mixed Mo | del for Repeated Measures for Change from Bas | seline in Total Score | (mITT Population) |
| Table 14.2.2.5.4 | : Linear Mixed Mo | del for Repeated Measures for Change from Bas | seline in Total Score | (PP Population) |
| Table 14.2.2.6.1 | Density: R | esults and Change from Baseline | | (mITT Population) |
| Table 14.2.2.6.2 | Density: L. 3, Visit 7 and End of Trea | near Mixed Model for Repeated Measures for Comment | hange from Baseline at Visit | (mITT Population) |
| Table 14.2.2.7.1 | Severe CCI | : Mean Annual Rate by Negative | Binomial Model | (mITT Population) |
| Table 14.2.2.7.2 | Time to ccl | Exacerbation: Kaplan-Meier Estir | nates | (mITT Population) |
| Table 14.2.2.8.1 | CCI | -cc Days: Summary Statistics | | (mITT Population) |
| Table 14.2.2.8.2 | CCI | CCI Days: ANCOVA model | | (mITT Population) |
| Table 14.2.2.9 | CCI | | | (mITT Population) |
| Table 14.2.2.10.1 | CCI | | | (mITT Population) |
| Table 14.2.2.10.2 | CCI | : Mean Annual Rate b | by Negative Binomial Model | (mITT Population) |
| Table 14.2.2.11.1 | CCI : Do | main Scores Results and Change Versus Baselin | ne | (mITT Population) |
| Table 14.2.2.11.2 | CCI : L | inear Mixed Model for Repeated Measures for | or Change from Baseline in | (mITT Population) |

# **5.3.4 Section 14.3: Safety**

| Table 14.3.1.1 | Summary of Treatment Emergent Adverse Events | (Safety Population) |
|---|---|---|
| Table 14.3.1.2.1 | Treatment Emergent Adverse Events by System Organ Class and Preferred Term | (Safety Population) |
| Table 14.3.1.2.2 | Serious Treatment Emergent Adverse Events by System Organ Class and Preferred Term | (Safety Population) |
| Table 14.3.1.2.3 | Related Treatment Emergent Adverse Events by System Organ Class and Preferred Term | (Safety Population) |
| Table 14.3.1.2.4 | Serious Related Treatment Emergent Adverse Events by System Organ Class and Preferred Term | (Safety Population) |
| Table 14.3.1.2.5 | Treatment Emergent Adverse Events Leading to Permanent IMP Discontinuation by System Organ Class and Preferred Term | (Safety Population) |
| Table 14.3.1.2.6 | Fatal Treatment Emergent Adverse Events by System Organ Class and Preferred Term | (Safety Population) |
| Table 14.3.1.3.1 | Treatment Emergent Adverse Events by System Organ Class, Preferred Term and Maximum Severity | (Safety Population) |

| Table 14.3.1.3.2 Related Treatment Emergent Adverse Events by System Organ Class, Preferred Term and Maximum Severity Most Frequent Treatment Emergent Adverse Events by Preferred Term (>=5% of Subjects with Events (Safety Population) in Any Group) Table 14.3.2.1 Listing of Adverse Events Leading to Death Table 14.3.2.2 Listing of Serious Adverse Events Leading to Discontinuation of Study Treatment Please Note: Section 14.3.3 (Narratives of Deaths, Other Serious and Certain Other Significant Adverse Events) is not to be used for any tables Spirometry: Felvy and FVC Results and Change Versus Baseline Table 14.3.4.1.1 Spirometry: Bronchospasm following IMP Administration at Visit 7 (End of Treatment) (Safety Population) Table 14.3.4.2.1 Vital Signs: Results and Change Versus Baseline (Safety Population) Table 14.3.4.2.2 Vital Signs: Stormal/Abnormal NCS/Abnormal CS Results (Safety Population) Table 14.3.4.2.3 Vital Signs: Shift Table (Safety Population) Table 14.3.4.3.1 Physical Examination: Results Physical Examination: Results Table 14.3.4.4.1 12-lead ECG: Results (Safety Population) Table 14.3.4.5.1.1 Haematology: Results and Change Versus Baseline (Safety Population) Table 14.3.4.5.1.1 Haematology: Results and Change Versus Baseline (Safety Population) Table 14.3.4.5.1.2 Haematology: Shift Table (Safety Population) Table 14.3.4.5.1.1 Haematology: Shift Table (Safety Population) Table 14.3.4.5.1.1 Haematology: Shift Table (Safety Population) Table 14.3.4.5.1.2 Clinical Chemistry: Shift Table (Safety Population) Table 14.3.4.6.1 Society (Clinical Chemistry: Shift Table (Safety Population) Table 14.3.4.6.1 Society (Clinical Chemistry: Shift Table (Safety Population) Table 14.3.4.6.1 Society (Safety Population) Table 14. | Sponsor: | Zambon S.p.A. | Protocol Number: | Z7224L02 | |
|---|---|---|---|---|---|
| Table 14.3.2.1 Listing of Adverse Events Leading to Death Listing of Serious Adverse Events Lable 14.3.2.2 Listing of Serious Adverse Events Lable 14.3.2.3 Listing of Adverse Events Leading to Discontinuation of Study Treatment Listing of Serious Adverse Events Leading to Discontinuation of Study Treatment Listing of Adverse Events Leading to Discontinuation of Study Treatment Listing of Adverse Events Leading to Discontinuation of Study Treatment Spirometry: FEV; and FVC Results and Change Certain Other Significant Adverse Events) is not to be used for any tables Spirometry: Bronchospasm following IMP Administration at Visit 7 (End of Treatment) Spirometry: Bronchospasm following IMP Administration at Visit 7 (End of Treatment) Vital Signs: Results and Change Versus Baseline (Safety Population) Table 14.3.4.2.1 Vital Signs: Shift Table (Safety Population) Table 14.3.4.3.1 Physical Examination: Results Table 14.3.4.3.1 Physical Examination: Results Table 14.3.4.4.1 12-lead ECG: Results (Safety Population) Table 14.3.4.5.1.1 (Safety Population) Table 14.3.4.5.1.1 (Safety Population) Table 14.3.4.5.1.1 (Safety Population) Table 14.3.4.5.1.2 (Safety Population) Table 14.3.4.5.1.2 (Safety Population) Table 14.3.4.5.1.1 (Safety Population) Table 14.3.4.5.1.2 (Safety Population) Table 14.3.4.5.1.2 (Safety Population) Table 14.3.4.5.1.1 (Safety Population) Table 14.3.4.5.1.2 (Safety Population) Table 14.3.4.5.1.2 (Safety Population) Table 14.3.4.5.1.2 (Safety Population) Table 14.3.4.6.1 (Safety Population) T | Table 14.3.1.3.2 | | s by System Organ Class, Preferred | Term and Maximum | (Safety Population) |
| Table 14.3.2.2 Listing of Serious Adverse Events Table 14.3.2.3 Listing of Adverse Events Leading to Discontinuation of Study Treatment Please Note: Section 14.3.3 (Narratives of Deaths, Other Serious and Certain Other Significant Adverse Events) is not to be used for any tables Spirometry: FEV1 and FVC Results and Change Versus Baseline Spirometry: Bronchospasm following IMP Administration at Visit 7 (End of Treatment) Spirometry: Bronchospasm following IMP Administration at Visit 7 (End of Treatment) Spirometry: Bronchospasm following IMP Administration at Visit 7 (End of Treatment) Spirometry: Bronchospasm following IMP Administration at Visit 7 (End of Treatment) Spirometry: Bronchospasm following IMP Administration at Visit 7 (End of Treatment) Safety Population) Vital Signs: Results and Change Versus Baseline Safety Population Table 14.3.4.2.1 Vital Signs: Normal/Abnormal NCS/Abnormal CS Results Safety Population Table 14.3.4.3.1 Physical Examination: Results Safety Population Physical Examination: Shift Table Safety Population Safety Population Table 14.3.4.4.1 12-lead ECG: Results Safety Population Table 14.3.4.5.1.1 Haematology: Results and Change Versus Baseline Safety Population Table 14.3.4.5.1.2 Haematology: Shift Table Safety Population Safety Population Table 14.3.4.5.1.1 Clinical Chemistry: Results and Change Versus Baseline Safety Population Table 14.3.4.5.1.1 Clinical Chemistry: Shift Table Safety Population Table 14.3.4.5.2.2 Clinical Chemistry: Shift Table Table 14.3.4.5.2.1 Clinical Chemistry: Shift Table Table 14.3.4.5.2.2 Clinical Chemistry: Shift Table Table 14.3.4.6.1 Safety Population Table 14.3.4.6.1 Safety Population Table 14.3.4.6.1 Safety Population Table 14.3.4.5.1 Safet | Table 14.3.1.4 | | Events by Preferred Term (>=5% or | f Subjects with Events | (Safety Population) |
| Table 14.3.2.3 Listing of Adverse Events Leading to Discontinuation of Study Treatment Please Note: Section 14.3.3 (Narratives of Deaths, Other Serious and Certain Other Significant Adverse Events) is not to be used for any tables Table 14.3.4.1.1 Spirometry: FEV1 and FVC Results and Change Versus Baseline (Safety Population) Table 14.3.4.2.1 Vital Signs: Results and Change Versus Baseline (Safety Population) Table 14.3.4.2.2 Vital Signs: Normal/Abnormal NCS/Abnormal CS Results Table 14.3.4.2.3 Vital Signs: Shift Table (Safety Population) Table 14.3.4.3.1 Physical Examination: Shift Table Table 14.3.4.3.2 Physical Examination: Shift Table Table 14.3.4.4.1 12-lead ECG: Results Table 14.3.4.4.1 12-lead ECG: Shift Table Table 14.3.4.5.1.1 Haematology: Results and Change Versus Baseline Table 14.3.4.5.1.2 Table 14.3.4.5.1.1 Haematology: Shift Table Table 14.3.4.5.1.2 Clinical Chemistry: Results and Change Versus Baseline Table 14.3.4.5.2.1 Clinical Chemistry: Results and Change Versus Baseline Table 14.3.4.5.2.1 Clinical Chemistry: Shift Table Table 14.3.4.5.2.2 Clinical Chemistry: Shift Table Table 14.3.4.6.1 Sodjum/Colistin) 5.4 Listing 16.1.7 Randomisation Listing 16.2.1.1 Subject Disposition Listing 16.2.2.1 Protocol Deviations – Analysis Populations | Table 14.3.2.1 | Listing of Adverse Events Leading to Death | | | |
| Please Note: Section 14.3.3 (Narratives of Deaths, Other Serious and Certain Other Significant Adverse Events) is not to be used for any tables Table 14.3.4.1.1 Spirometry: FFV <sub>1</sub> and FVC Results and Change Versus Baseline (Safety Population) Table 14.3.4.2.1 Vital Signs: Results and Change Versus Baseline (Safety Population) Table 14.3.4.2.2 Vital Signs: Normal/Abnormal NCS/Abnormal CS Results (Safety Population) Table 14.3.4.2.3 Vital Signs: Normal/Abnormal NCS/Abnormal CS Results (Safety Population) Table 14.3.4.3.1 Physical Examination: Results (Safety Population) Table 14.3.4.3.2 Physical Examination: Results (Safety Population) Table 14.3.4.4.1 12-lead ECG: Results (Safety Population) Table 14.3.4.4.2 12-lead ECG: Shift Table (Safety Population) Table 14.3.4.5.1.1 Haematology: Results and Change Versus Baseline (Safety Population) Table 14.3.4.5.1.2 Haematology: Shift Table (Safety Population) Table 14.3.4.5.1.2 Haematology: Shift Table (Safety Population) Table 14.3.4.5.2.1 Clinical Chemistry: Results and Change Versus Baseline (Safety Population) Table 14.3.4.5.2.2 Clinical Chemistry: Results and Change Versus Baseline (Safety Population) Table 14.3.4.6.1 Sodium/Colistin) Table 14.3.4.6.1 Sodium/Colistin) Table 14.3.4.6.2 Randomisation Listing 16.1.7 Randomisation Listing 16.2.1.1 Subject Disposition Listing 16.2.2.1 Protocol Deviations – Analysis Populations | Table 14.3.2.2 | | | | |
| Table 14.3.4.1.1 Spirometry: FEV1 and FVC Results and Change Versus Baseline (Safety Population) Spirometry: Bronchospasm following IMP Administration at Visit 7 (End of Treatment) (Safety Population) Vital Signs: Results and Change Versus Baseline (Safety Population) Vital Signs: Normal/Abnormal NCS/Abnormal CS Results (Safety Population) Vital Signs: Shift Table (Safety Population) Vital Signs: Shift Table (Safety Population) Vital Signs: Shift Table (Safety Population) Physical Examination: Results (Safety Population) Physical Examination: Shift Table (Safety Population) Physical Examination: Shift Table (Safety Population) Physical Examination: Shift Table (Safety Population) 12-lead ECG: Results (Safety Population) 12-lead ECG: Shift Table (Safety Population) 12-lead ECG | | | | | |
| Table 14.3.4.1.2 Spiromety: Bronchospasm following IMP Administration at Visit 7 (End of Treatment) (Safety Population) Table 14.3.4.2.1 Vital Signs: Results and Change Versus Baseline (Safety Population) Vital Signs: Normal/Abnormal NCS/Abnormal CS Results Table 14.3.4.2.2 Vital Signs: Shift Table (Safety Population) Table 14.3.4.3.1 Physical Examination: Results (Safety Population) Table 14.3.4.3.2 Physical Examination: Shift Table (Safety Population) Table 14.3.4.4.1 12-lead ECG: Results (Safety Population) Table 14.3.4.5.1.1 Haematology: Results and Change Versus Baseline (Safety Population) Table 14.3.4.5.1.2 Clinical Chemistry: Results and Change Versus Baseline (Safety Population) Table 14.3.4.5.2.1 Clinical Chemistry: Results and Change Versus Baseline (Safety Population) Table 14.3.4.5.2.2 Clinical Chemistry: Results and Change Versus Baseline (Safety Population) Table 14.3.4.6.1 Clinical Chemistry: Shift Table (Safety Population) Table 14.3.4.6.1 Clinical Chemistry: Shift Table (Safety Population) Table 14.3.4.6.2 Clinical Chemistry: Shift Table (Safety Population) Table 14.3.4.6.2 Clinical Chemistry: Shift Table (Safety Population) Table 14.3.4.6.1 Sodium/Colistin) Table 14.3.4.6.2 Clinical Chemistry: Shift Table (Safety Population) Table 14.3.4.6.2 Clinical Chemistry: Shift Table (Safety Population) Table 14.3.4.6.2 Sodium/Colistin) Table 14.3.4.6.2 Sodium/Colistin (Last Available Data) (Overall and by Previous Use of Colistimethate Sodium/Colistin) 5.4 Listing 16.1.7 Randomisation Listing 16.2.1.1 Subject Disposition Protocol Deviations – Analysis Populations Protocol Deviations – Analysis Populations | Please Note: Section | 14.3.3 (Narratives of Deaths, Other Serious and Ce | ertain Other Significant Adverse Eve | nts) is not to be used for | or any tables |
| Table 14.3.4.2.1 Vital Signs: Results and Change Versus Baseline Table 14.3.4.2.2 Vital Signs: Normal/Abnormal NCS/Abnormal CS Results Table 14.3.4.2.3 Vital Signs: Shift Table Table 14.3.4.3.1 Physical Examination: Results Table 14.3.4.3.2 Physical Examination: Shift Table Table 14.3.4.4.1 12-lead ECG: Results Table 14.3.4.4.1 12-lead ECG: Shift Table Table 14.3.4.5.1.1 Haematology: Results and Change Versus Baseline Table 14.3.4.5.1.2 Table 14.3.4.5.1.2 Haematology: Shift Table Table 14.3.4.5.2.1 Clinical Chemistry: Results and Change Versus Baseline Table 14.3.4.5.2.2 Clinical Chemistry: Results and Change Versus Baseline Table 14.3.4.6.1 Sodium/Colistin) Table 14.3.4.6.2 Sodium/Colistin) Table 14.3.4.6.2 Table Listing 16.1.7 Randomisation Listing 16.2.1.1 Subject Disposition Listing 16.2.2.1 Protocol Deviations – Analysis Populations Listing 16.2.2.1 Protocol Deviations – Analysis Populations | Table 14.3.4.1.1 | 1 | | | (Safety Population) |
| Table 14.3.4.2.2 Vital Signs: Normal/Abnormal NCS/Abnormal CS Results Table 14.3.4.2.3 Vital Signs: Shift Table (Safety Population) Physical Examination: Results (Safety Population) Physical Examination: Shift Table (Safety Population) Physical Examination: Shift Table (Safety Population) Table 14.3.4.3.1 Physical Examination: Shift Table (Safety Population) Table 14.3.4.4.1 12-lead ECG: Results (Safety Population) Table 14.3.4.5.1.1 Haematology: Results and Change Versus Baseline Table 14.3.4.5.1.1 Haematology: Shift Table (Safety Population) Table 14.3.4.5.1.2 Clinical Chemistry: Results and Change Versus Baseline (Safety Population) Table 14.3.4.5.2.1 Clinical Chemistry: Results and Change Versus Baseline (Safety Population) Table 14.3.4.6.1 Sodium/Colistin) Table 14.3.4.6.1 Colistimethate Sodium/Colistin) Table 14.3.4.6.2 Colistimethate Sodium/Colistin) Table 14.3.4.6.1 Subject Disposition Listing 16.2.1.1 Subject Disposition Listing 16.2.2.1 Protocol Deviations – Analysis Populations | Table 14.3.4.1.2 | | | tment) | |
| Table 14.3.4.2.3 Vital Signs: Shift Table Table 14.3.4.3.1 Physical Examination: Results Table 14.3.4.3.2 Physical Examination: Shift Table Table 14.3.4.3.1 Physical Examination: Shift Table Table 14.3.4.3.1 12-lead ECG: Results Table 14.3.4.3.1 12-lead ECG: Shift Table Table 14.3.4.5.1.1 Haematology: Results and Change Versus Baseline Table 14.3.4.5.1.2 Haematology: Shift Table Table 14.3.4.5.1.1 Clinical Chemistry: Results and Change Versus Baseline Table 14.3.4.5.2.1 Clinical Chemistry: Results and Change Versus Baseline Table 14.3.4.5.2.2 Clinical Chemistry: Shift Table Table 14.3.4.6.1 Colinical | | | | | |
| Table 14.3.4.3.1 Physical Examination: Results Population) Table 14.3.4.3.2 Physical Examination: Shift Table Table 14.3.4.3.2 Physical Examination: Shift Table Table 14.3.4.4.1 12-lead ECG: Results (Safety Population) Table 14.3.4.4.2 12-lead ECG: Shift Table Table 14.3.4.5.1.1 Haematology: Results and Change Versus Baseline Table 14.3.4.5.1.2 Haematology: Shift Table Table 14.3.4.5.2.1 Clinical Chemistry: Results and Change Versus Baseline Table 14.3.4.5.2.2 Clinical Chemistry: Results and Change Versus Baseline Table 14.3.4.6.1 Clinical Chemistry: Shift Table Table 1 | | | al CS Results | | |
| Table 14.3.4.3.2 Physical Examination: Shift Table Table 14.3.4.4.1 12-lead ECG: Results Table 14.3.4.4.2 12-lead ECG: Shift Table Table 14.3.4.5.1.1 Haematology: Results and Change Versus Baseline Table 14.3.4.5.1.2 (Safety Population) Table 14.3.4.5.2.1 Clinical Chemistry: Results and Change Versus Baseline Table 14.3.4.5.2.1 Clinical Chemistry: Shift Table Table 14.3.4.5.2.2 Clinical Chemistry: Shift Table Table 14.3.4.6.1 Sodium/Colistin) Table 14.3.4.6.1 Colistimethate Table 14.3.4.6.1 Sodium/Colistin) Table 14.3.4.6.2 Colistimethate Sodium/Colistin) Listing 16.1.7 Randomisation Listing 16.2.1.1 Subject Disposition Listing 16.2.2.1 Protocol Deviations – Analysis Populations | Table 14.3.4.2.3 | | | | |
| Table 14.3.4.4.1 Table 14.3.4.4.2 Table 14.3.4.5.1.1 Table 14.3.4.5.1.1 Table 14.3.4.5.1.1 Table 14.3.4.5.1.2 Table 14.3.4.5.2.1 Table 14.3.4.5.2.1 Table 14.3.4.5.2.1 Table 14.3.4.5.2.2 Table 14.3.4.5.2.2 Table 14.3.4.5.2.2 Table 14.3.4.5.3.3 Table 14.3.4.5.3 Table 14.3.4.5 Ta | | • | | | |
| Table 14.3.4.4.2 Table 14.3.4.4.2 Table 14.3.4.5.1.1 Table 14.3.4.5.1.1 Haematology: Results and Change Versus Baseline Table 14.3.4.5.1.2 Haematology: Shift Table Table 14.3.4.5.2.1 Clinical Chemistry: Results and Change Versus Baseline Table 14.3.4.5.2.2 Clinical Chemistry: Shift Table Table 14.3.4.6.1 Table 14.3.4.6.1 Table 14.3.4.6.1 Table 14.3.4.6.2 Collimical Chemistry: Shift Table Collimical Chemistry: Shift Table (Safety Population) (Safety Population) (Safety Population) Table 14.3.4.6.2 Collimical Chemistry: Shift Table (Safety Population) (Safety Population) (Safety Population) (Safety Population) Table 14.3.4.6.2 Collimical Chemistry: Shift Table (Safety Population) (Safety Population) (Safety Population) Table 14.3.4.6.1 Table 14.3.4.6.2 Collimical Chemistry: Shift Table (Safety Population) (Safety Population) (Safety Population) Table 14.3.4.6.2 Table 14.3.4.6.1 Sodium/Colistin) Table 14.3.4.6.1 Table 14.3.4.6.1 Sodium/Colistin) Table 14.3.4.6.1 Table 14.3.4.6. | Table 14.3.4.3.2 | Physical Examination: Shift Table | | | (Safety Population) |
| Table 14.3.4.5.1.1 Haematology: Results and Change Versus Baseline Table 14.3.4.5.1.2 Haematology: Shift Table Table 14.3.4.5.2.1 Clinical Chemistry: Results and Change Versus Baseline Table 14.3.4.5.2.2 Clinical Chemistry: Shift Table Table 14.3.4.6.1 Clinical Chemistry: Shift Table Table 14.3.4.6.1 Sodium/Colistin) Table 14.3.4.6.2 Clinical Chemistry: Shift Table CCI Sodium/Colistin) (Safety Population) Table 14.3.4.6.2 Colistimethate Sodium/Colistin) 5.4 Listings Listing 16.1.7 Randomisation Subject Disposition Listing 16.2.1.1 Subject Disposition Protocol Deviations – Analysis Populations | Table 14.3.4.4.1 | 12-lead ECG: Results | | | (Safety Population) |
| Table 14.3.4.5.1.2 Haematology: Shift Table Table 14.3.4.5.2.1 Clinical Chemistry: Results and Change Versus Baseline Clinical Chemistry: Shift Table Clinical Chemistry: Shift Table Clinical Chemistry: Shift Table Table 14.3.4.5.2.2 Clinical Chemistry: Shift Table Table 14.3.4.6.1 Sodium/Colistin) Table 14.3.4.6.2 Colistimethate Sodium/Colistin) Table 14.3.4.6.2 Colistimethate Sodium/Colistin) Listing 16.1.7 Randomisation Listing 16.2.1.1 Subject Disposition Listing 16.2.2.1 Protocol Deviations – Analysis Populations | | | | | |
| Table 14.3.4.5.2.1 Clinical Chemistry: Results and Change Versus Baseline Table 14.3.4.5.2.2 Clinical Chemistry: Results and Change Versus Baseline Clinical Chemistry: Shift Table Table 14.3.4.6.1 Sodium/Colistin Table 14.3.4.6.2 Colistimethate Sodium/Colistin Listing 16.1.7 Listing 16.2.1.1 Listing 16.2.2.1 Protocol Deviations – Analysis Populations Clinical Chemistry: Results and Change Versus Baseline (Safety Population) (Safety Population) (Safety Population) (Safety Population) (Safety Population) Clast Available Data) (Overall and by Previous Use of Safety Population) | Table 14.3.4.5.1.1 | · | seline | | |
| Table 14.3.4.5.2.2 Clinical Chemistry: Shift Table Table 14.3.4.6.1 Sodium/Colistin) Table 14.3.4.6.2 Clinical Chemistry: Shift Table Sodium/Colistin) (Safety Population) | | | | | |
| Table 14.3.4.6.1 Sodium/Colistin) Table 14.3.4.6.2 Colistimethate Sodium/Colistin) Listing 16.1.7 Listing 16.2.1.1 Listing 16.2.2.1 Protocol Deviations — Analysis Populations at Visit 7 (Overall and by Previous Use of Colistimethate (Safety Population) (Last Available Data) (Overall and by Previous Use of (Safety Population) | | | sus Baseline | | |
| Table 14.3.4.6.1 Sodium/Colistin) Table 14.3.4.6.2 Sodium/Colistin) (Last Available Data) (Overall and by Previous Use of Colistimethate Sodium/Colistin) Listing 16.1.7 Randomisation Listing 16.2.1.1 Subject Disposition Listing 16.2.2.1 Protocol Deviations – Analysis Populations | Table 14.3.4.5.2.2 | • | | | (Safety Population) |
| Colistimethate Sodium/Colistin) 5.4 Listings Listing 16.1.7 Randomisation Listing 16.2.1.1 Subject Disposition Listing 16.2.2.1 Protocol Deviations – Analysis Populations | Table 14.3.4.6.1 | | Visit 7 (Overall and by Previous 1 | Use of Colistimethate | (Safety Population) |
| Listing 16.1.7 Randomisation Listing 16.2.1.1 Subject Disposition Listing 16.2.2.1 Protocol Deviations – Analysis Populations | Table 14.3.4.6.2 | | Last Available Data) (Overall and | by Previous Use of | (Safety Population) |
| Listing 16.2.1.1 Subject Disposition Listing 16.2.2.1 Protocol Deviations – Analysis Populations | 5.4 Listings | | | | |
| Listing 16.2.2.1 Protocol Deviations – Analysis Populations | | | | | |
| • 1 | | | | | |
| Listing 16.2.3.1 Inclusion Criteria | _ | | | | |
| | Listing 16.2.3.1 | Inclusion Criteria | | | |

Z7224L02

| Sponsor: | Zambon S.p.A. | Protocol Number: | |
|---|---|---|--|
| Listing 16.2.3.2 | Violations to Inclusion Criteria | | |
| Listing 16.2.3.3 | Exclusion Criteria | | |
| Listing 16.2.3.4 | Violations to Exclusion Criteria | | |
| Listing 16.2.4.1 | Subject Demography | | |
| Listing 16.2.4.2 | Smoking / Alcohol Status | | |
| Listing 16.2.4.3 | Medical History | | |
| Listing 16.2.4.4 | Non-CF Bronchiectasis History | | |
| Listing 16.2.4.5 | Prior and Concomitant Medications | | |
| Listing 16.2.4.6 | Systemic Antibiotic Therapy | | |
| Listing 16.2.5.1.1 | IMP Administration under Clinical Supervis | sion and Training on IMP Preparation | |
| Listing 16.2.5.1.2 | IMP and Salbutamol/Albuterol Dispensing | | |
| Listing 16.2.5.2.1 | Dispensing, Training, Collection and | Status | |
| Listing 16.2.5.2.2 | <b>CCI</b> Data | | |
| Listing 16.2.5.3 | Exposure and Adherence | | |
| Listing 16.2.6 | Visit Dates | | |
| Listing 16.2.7.1 | Adverse Events | | |
| Listing 16.2.7.2 | Related Adverse Events | | |
| Listing 16.2.7.3 | Severe Adverse Events | | |
| Listing 16.2.7.4.1 | NCFB Pulmonary Exacerbation: eCRF Data | | |
| Listing 16.2.7.4.2 | NCFB Pulmonary Exacerbation: Derived D | ata | |
| Listing 16.2.8.1 | 12-Lead ECG | | |
| Listing 16.2.8.2.1 | Haematology | | |
| Listing 16.2.8.2.2 | Clinial Chemistry | | |
| Listing 16.2.8.3 | Vital Signs | | |
| Listing 16.2.8.4 | Physical Examination | | |
| Listing 16.2.8.5 | Pregnancy Test (Urine Dipstick) | | |
| Listing 16.2.8.6 | Spirometry: FEV <sub>1</sub> and FVC | | |
| Listing 16.2.8.7 | Collection and Results | | |
| Listing 16.2.8.8 | CCI | | |
| Listing 16.2.8.9 | CCI CCI | | |
| Sponsor: | Zambon S.p.A. | Protocol Number: | Z7224L02 |
|----------|---------------|------------------|----------|
| • | • | | |

### 5.5 Figures

| Figure 14.2.1.1.11 | Forest Plot for Rate Ratio (Colistimethate Sodium versus Placebo) | of NCFB Pulmonary | (mITT Population) |
|---|---|---|---|
| | Exacerbations by Subgroup | | |
| Figure 14.2.2.1.3 | Kaplan-Meier Curve for CCI | | (mITT Population) |
| Figure 14.2.2.1.4 | Kaplan-Meier Curve for CCI | | (PP Population) |
| Figure 14.2.2.5.5 | Change from Baseline in CCI by Visit | | (mITT Population) |
| Figure 14.2.2.6.3 | Change from Baseline in CCI by Visit | | (mITT Population) |

Tables, Listings, and Figures will follow the format of: Zambon-Z7224L02-SAP-Shells-FINAL-v2.0-dd-Mmm-yyyy; where dd-Mmm-yyyy denotes the date of the Final v2.0 shells document.

| Sponsor: Zambon S.p.A. | Protocol Number: | Z7224L02 |
|------------------------|------------------|----------|
|------------------------|------------------|----------|

#### 5.6 References

- 1 Keene, O. N., Roger, J. H., Hartley, B. F. and Kenward, M. G. (2014), Missing data CCI for recurrent event data using controlled imputation. Pharmaceut. Statist., 13: 258-264. doi:10.1002/pst.1624
- 2 Barnard J, Rubin D. Small-sample degrees of freedom with multiple imputation. Biometrika 1999; 86:948–955.
- 3 Leila DAF Amorim, Jianwen Cai; Modelling recurrent events: a tutorial for analysis in epidemiology, International Journal of Epidemiology, Volume 44, Issue 1, 1 February 2015, Pages 324–333, https://doi.org/10.1093/ije/dyu222
- 4 Koch, G. G., Tangen, C. M., Jung, J. and Amara, I. A. (1998), Issues for covariance analysis of dichotomous and ordered categorical data from randomized clinical trials and non- parametric strategies for addressing them. Statist. Med., 17: 1863-1892. doi:10.1002/(SICI)1097-0258(19980815/30)17:15/16<1863::AID-SIM989>3.0.CO;2-M
- 5 Dmitrienko A, Molenberghs G, Chuang-Stein C, Offen W; Analysis of Clinical Trials Using SAS: A Practical Guide. Cary, NC: SAS Press; 2007.
- 6 Satterthwaite, F. W. (1946), An Approximate Distribution of Estimates of Variance Components, Biometrics Bulletin, 2, 110–114.
- Appendix 1 to the CHMP guideline on the evaluation of anticancer medicinal products in man (EMEA/CHMP/EWP/27994/2008).
- Bronchiectasis manual. Previously available from: http://www.psy.miami.edu/qol b/scoring.phtml
- , Version 2.3. Division of Cardiac and Vascular Science, Col., University of London.
- 10 Quanjer et al., Multi-ethnic reference values for spirometry for the 3-95-yr age range: the global lung function 2012 equations, Eur Respir J. 2012 Dec 40(6):1324-43.

| Sponsor: | Zambon S.p.A. | Protocol Number: | Z7224L02 |
|-----------------|---------------|------------------|----------|
| Appendix 1: CCI | | | |

Below weights for each item and other details for

calculation are reported.

Please tick in one box to show how you describe your current health (not used in total or domain score calculations):

| Response |
|-----------|
| Very good |
| Good |
| Fair |
| Poor |
| Very poor |

#### **ITEM WEIGHTS**

#### PART 1

1) Over the past 4 weeks / 3 months, I have coughed:

| Response | Weight |
|----------------------------|--------|
| Most days a week | 80.6 |
| Several days a week | 63.2 |
| A few days a month | 29.3 |
| Only with chest infections | 28.1 |
| Not at all | 0.0 |

2) Over the past 4 weeks / 3 months, I have brought up phlegm (sputum):

| Response | Weight |
|----------------------------|--------|
| Most days a week | 76.8 |
| Several days a week | 60.0 |
| A few days a month | 34.0 |
| Only with chest infections | 30.2 |
| Not at all | 0.0 |

3) Over the past 4 weeks / 3 months, I have had shortness of breath:

| Response | Weight |
|----------------------------|--------|
| Most days a week | 87.2 |
| Several days a week | 71.4 |
| A few days a month | 43.7 |
| Only with chest infections | 35.7 |
| Not at all | 0.0 |

# 4) Over the past 4 weeks / 3 months, I have had attacks of wheezing: Response Weight

| Sponsor: | Zambon S.p.A. | | Protocol Number: | Z7224L02 |
|---|---|---|---|---|
| Most days a w<br>Several days a | ı week | 86.2<br>71.0 | | |
| A few days a | | 45.6 | | |
| Only with che | est infections | 36.4 | | |
| Not at all | | 0.0 | | |

5) During the past 4 weeks / 3 months, how many severe or very unpleasant attacks of chest trouble have you had?

| Response | Weight |
|-------------------------|--------|
| More than three attacks | 86.7 |
| 3 attacks | 73.5 |
| 2 attacks | 60.3 |
| 1 attack | 44.2 |
| No attacks | 0.0 |

6) How long did the worst attack of chest trouble last?

| Response | Weight |
|-----------------|--------|
| A week or more | 89.7 |
| 3 or more days | 73.5 |
| 1 or 2 days | 58.8 |
| Less than a day | 41.9 |

7) Over the past 4 weeks / 3 months, in an average week, how many good days (with little chest trouble) have you had?

| Response | Weight |
|--------------------------|--------|
| No good days | 93.3 |
| 1 or 2 good days | 76.6 |
| 3 or 4 good days | 61.5 |
| Nearly every day is good | 15.4 |
| Every day is good | 0.0 |

8) If you have a wheeze, is it worse in the morning?

| Response | Weight |
|----------|--------|
| No | 0.0 |
| Yes | 62.0 |

#### PART 2

#### Section 1

How would you describe your chest condition?

| Response | Weight |
|-----------------------------------|--------|
| The most important problem I have | 83.2 |
| Causes me quite a lot of problems | 82.5 |
| Causes me a few problems | 34.6 |
| Causes no problem | 0.0 |

#### If you have ever had paid employment.

| Response | Weight |
|--------------------------------------------------------------------|--------|
| My chest trouble made me stop work altogether | 88.9 |
| My chest trouble interferes with my work or made me change my work | 77.6 |
| My chest trouble does not affect my work | 0.0 |

#### Section 2

Questions about what activities usually make you feel breathless these days.

| Response | Weight |
|-------------------------------|--------|
| Sitting or lying still | 90.6 |
| Getting washed or dressed | 82.8 |
| Walking around the home | 80.2 |
| Walking outside on the level | 81.4 |
| Walking up a flight of stairs | 76.1 |
| Walking up hills | 75.1 |
| Playing sports or games | 72.1 |

#### Section 3

Some more questions about your cough and breathlessness these days.

| Response | Weight |
|-----------------------------------------|--------|
| My cough hurts | 81.1 |
| My cough makes me tired | 79.1 |
| I am breathless when I talk | 84.5 |
| I am breathless when I bend over | 76.8 |
| My cough or breathing disturbs my sleep | 87.9 |
| I get exhausted easily | 84.0 |

#### **Section 4**

Questions about other effects that your chest trouble may have on you these days.

| Response | Weight |
|--------------------------------------------------------------------|--------|
| My cough or breathing is embarrassing in public | 74.1 |
| My chest trouble is a nuisance to my family, friends or neighbours | 79.1 |
| I get afraid or panic when I cannot get my breath | 87.7 |
| I feel that I am not in control of my chest problem | 90.1 |
| I do not expect my chest to get any better | 82.3 |
| I have become frail or an invalid because of my chest | 89.9 |
| Exercise is not safe for me | 75.7 |
| Everything seems too much of an effort | 84.5 |

#### Section 5

# Questions about your medication, if you are receiving no medication go straight to section 6.

| Response | Weight |
|---------------------------------------------------|--------|
| My medication does not help me very much | 88.2 |
| I get embarrassed using my medication in public | 53.9 |
| I have unpleasant side effects from my medication | 81.1 |
| My medication interferes with my life a lot | 70.3 |

| Sponsor: Zambon S.p.A. Protocol Nun | nber: Z7224L02 |
|-------------------------------------|----------------|
|-------------------------------------|----------------|

#### Section 6

#### These are questions about how your activities might be affected by your breathing.

| Response | Weight |
|---|---|
| I take a long time to get washed or dressed | 74.2 |
| I cannot take a bath or shower, or I take a long time | 81.0 |
| I walk slower than other people, or I stop for rests | 71.7 |
| Jobs such as housework take a long time, or I have to stop for rests | 70.6 |
| If I walk up one flight of stairs, I have to go slowly or stop | 71.6 |
| If I hurry or walk fast, I have to stop or slow down | 72.3 |
| My breathing makes it difficult to do things such as walk up hills, carrying things | 74.5 |
| up stairs, light gardening such as weeding, dance, play bowls or play golf | |
| My breathing makes it difficult to do things such as carry heavy loads, dig the | 71.4 |
| garden or shovel snow, jog or walk at 5 miles per hour, play tennis or swim | |
| My breathing makes it difficult to do things such as very heavy manual work, run, | 63.5 |
| cycle, swim fast or play competitive sports | |

#### Section 7

We would like to know how your chest usually affects your daily life.

| Response | Weight |
|-------------------------------------------------|--------|
| I cannot play sports or games | 64.8 |
| I cannot go out for entertainment or recreation | 79.8 |
| I cannot go out of the house to do the shopping | 81.0 |
| I cannot do housework | 79.1 |
| I cannot move far from my bed or chair | 94.0 |

Please write in any other important activities that your chest trouble may stop you doing (not used in total or domain score calculations):

Now would you tick in the box (one only) which you think best describes how your chest affects you:

| Response | Weight |
|---------------------------------------------------------|--------|
| It does not stop me doing anything I would like to do | 0.0 |
| It stops me doing one or two things I would like to do | 42.0 |
| It stops me doing most of the things I would like to do | 84.2 |
| It stops me doing everything I would like to do | 96.7 |

#### **Scoring Algorithm**

Three domain scores are calculated: Symptoms, Activity, Impacts.

One Total score is also calculated.

| Sponsor: Zambon S.p.A. | Protocol Number: | Z7224L02 |
|------------------------|------------------|----------|
|------------------------|------------------|----------|

#### PRINCIPLE OF CALCULATION

Each questionnaire response (except where indicated) has a unique empirically derived 'weight'. The lowest possible weight is zero and the highest is 100.

#### Each domain of the questionnaire is scored separately in three steps:

- i. The weights for all items with positive responses are summed.
- ii The weights for missed items are deducted from the maximum possible weight for each domain. The weights for all missed items are deducted from the maximum possible weight for the Total score.
- iii. The score is calculated by dividing the summed weights by the adjusted maximum possible weight for that domain and expressing the result as a percentage:

$$Score = \frac{Summed weights from positive items in that domain}{Sum of weights for all items in that domain} *100$$

#### The Total score is calculated in similar way:

$$Score = \frac{Summed weights from positive items in the questionnaire}{Sum of weights for all items in the questionnaire} *100$$

#### Sum of maximum possible weights for each domain and Total:

| Symptoms | 662.5 |
|----------|--------|
| Activity | 1209.1 |
| Impacts | 2117.8 |
| Total | 3989.4 |

(Note: these are the maximum possible weights that could be obtained for the worst possible state of the subject).

#### SYMPTOMS DOMAIN

This is calculated from the summed weights for the positive responses to questions 1-8 of Part 1.

#### ACTIVITY DOMAIN

This is calculated from the summed weights for the positive responses to sections 2 and 6 of Part 2.

#### IMPACTS DOMAIN

This is calculated from the summed weights for the positive responses to sections 1, 3, 4, 5, 7 of Part 2.

#### TOTAL SCORE

The Total score is calculated by summing all positive responses in the questionnaire and expressing the result as a percentage of the total weight for the questionnaire.

#### HANDLING MISSING ITEMS

The following methods will be used:

#### **Symptoms**

The Symptoms domain will tolerate a maximum of 2 missed items. The weight for the missed item is subtracted from the total possible weight for the Symptoms domain (662.5) and from the Total weight (3989.4).

#### Activity

The Activity domain will tolerate a maximum of 4 missed items. The weight for the missed item is subtracted from the total possible weight for the Activity domain (1209.1) and from the Total weight (3989.4).

#### **Impacts**

The Impacts domain will tolerate a maximum of 6 missed items. The weight for the missed item is subtracted from the total possible weight for the Impacts domain (2117.8) and from the Total weight (3989.4).

### **Appendix 2: CCI**

CC

Below scores for each item and other details for calculation are reported.

The values assigned to participants' responses for each question are listed below.

#### 1) Performing vigorous activities, such as gardening or exercising

| Response | Score |
|---------------------|-------|
| A lot of difficulty | 1 |
| Moderate difficulty | 2 |
| A little difficulty | 3 |
| No difficulty | 4 |

#### 2) Walking as fast as others (family, friends, etc.)

| Response | Score |
|---------------------|-------|
| A lot of difficulty | 1 |
| Moderate difficulty | 2 |
| A little difficulty | 3 |
| No difficulty | 4 |

#### 3) Carrying heavy things, such as books or shopping bags.

| Response | Score |
|---------------------|-------|
| A lot of difficulty | 1 |
| Moderate difficulty | 2 |
| A little difficulty | 3 |
| No difficulty | 4 |

#### 4) Climbing one flight of stairs.

| Response | Score |
|---------------------|-------|
| A lot of difficulty | 1 |
| Moderate difficulty | 2 |
| A little difficulty | 3 |
| No difficulty | 4 |

#### 5) You felt well.

| Response | Score | Reverse-coded Score |
|-----------|-------|---------------------|
| Always | 1 | 4 |
| Often | 2 | 3 |
| Sometimes | 3 | 2 |
| Never | 4 | 1 |

#### 6) You felt tired.

| Response | Score |
|-----------|-------|
| Always | 1 |
| Often | 2 |
| Sometimes | 3 |
| Never | 4 |

#### 7) You felt anxious.

| Response | Score |
|-----------|-------|
| Always | 1 |
| Often | 2 |
| Sometimes | 3 |
| Never | 4 |

#### 8) You felt energetic.

| Response | Score | Reverse-coded Score |
|-----------|-------|---------------------|
| Always | 1 | 4 |
| Often | 2 | 3 |
| Sometimes | 3 | 2 |
| Never | 4 | 1 |

#### 9) You felt exhausted.

| Response | Score |
|-----------|-------|
| Always | 1 |
| Often | 2 |
| Sometimes | 3 |
| Never | 4 |

#### 10) You felt sad.

| Response | Score |
|-----------|-------|
| Always | 1 |
| Often | 2 |
| Sometimes | 3 |
| Never | 4 |

#### 11) You felt depressed.

| Response | Score |
|-----------|-------|
| Always | 1 |
| Often | 2 |
| Sometimes | 3 |
| Never | 4 |

| Sponsor: Zambon S.p.A. | Protocol Number: | Z7224L02 |
|------------------------|------------------|----------|
|------------------------|------------------|----------|

### 12) To what extent do your treatments for bronchiectasis make your daily life more difficult?

| Response | Score | Reverse-coded Score |
|------------|-------|---------------------|
| Not at all | 1 | 4 |
| A little | 2 | 3 |
| Moderately | 3 | 2 |
| A lot | 4 | 1 |

### 13) How much time do you currently spend each day on your treatments for bronchiectasis?

| Response | Score |
|-------------------|-------|
| A lot | 1 |
| A moderate amount | 2 |
| A little | 3 |
| Almost none | 4 |

#### 14) How difficult is it for you to fit in your treatments for bronchiectasis each day?

| Response | Score | Reverse-coded Score |
|------------|-------|---------------------|
| Not at all | 1 | 4 |
| A little | 2 | 3 |
| Moderately | 3 | 2 |
| Very | 4 | 1 |

#### 15) How do you think your health is now?

| Response | Score | Reverse-coded Score |
|-----------|-------|---------------------|
| Excellent | 1 | 4 |
| Good | 2 | 3 |
| Fair | 3 | 2 |
| Poor | 4 | 1 |

#### 16) I have to limit vigorous activities, such as walking or exercising

| Response | Score |
|-----------------|-------|
| Completely true | 1 |
| Mostly true | 2 |
| A little true | 3 |
| Not at all true | 4 |

#### 17) I have to stay at home more than I want to

| | Score |
|-------|-------|
| ponse | |

| Sponsor: Zambon S.p.A. Protocol Number: Z722 | '224L02 |
|----------------------------------------------|---------|
|----------------------------------------------|---------|

Completely true 1 Mostly true 2 A little true 3 Not at all true 4

#### 18) I am worried about being exposed to other people who are ill

| Response | Score |
|-----------------|-------|
| Completely true | 1 |
| Mostly true | 2 |
| A little true | 3 |
| Not at all true | 4 |

#### 19) It is difficult to be intimate with a partner (kissing, hugging, etc)

| Response | Score |
|-----------------|-------|
| Completely true | 1 |
| Mostly true | 2 |
| A little true | 3 |
| Not at all true | 4 |

#### 20) I lead a normal life

| Response | Score | Reverse-coded Score |
|-----------------|-------|---------------------|
| Completely true | 1 | 4 |
| Mostly true | 2 | 3 |
| A little true | 3 | 2 |
| Not at all true | 4 | 1 |

#### 21) I am concerned that my health will get worse

| Response | Score |
|-----------------|-------|
| Completely true | 1 |
| Mostly true | 2 |
| A little true | 3 |
| Not at all true | 4 |

#### 22) I think my coughing bothers other people

| Response | Score |
|-----------------|-------|
| Completely true | 1 |
| Mostly true | 2 |
| A little true | 3 |
| Not at all true | 4 |

#### 23) I often feel lonely

Response Score

| Sponsor: Zambon S.p.A. | Protocol Number: | Z7224L02 |
|------------------------|------------------|----------|
|------------------------|------------------|----------|

Completely true 1 Mostly true 2 A little true 3 Not at all true 4

#### 24) I feel healthy

| Response | Score | Reverse-coded Score |
|-----------------|-------|---------------------|
| Completely true | 1 | 4 |
| Mostly true | 2 | 3 |
| A little true | 3 | 2 |
| Not at all true | 4 | 1 |

#### 25) It is difficult to make plans for the future (holidays, attending family events, etc.)

| Response | Score |
|-----------------|-------|
| Completely true | 1 |
| Mostly true | 2 |
| A little true | 3 |
| Not at all true | 4 |

#### 26) I feel embarrassed when I am coughing

| Response | Score |
|-----------------|-------|
| Completely true | 1 |
| Mostly true | 2 |
| A little true | 3 |
| Not at all true | 4 |

### 27) To what extent did you have trouble keeping up with your job, housework, or other daily activities?

| Response | Score | Reverse-coded Score |
|---|---|---|
| You have had no trouble keeping up | 1 | 4 |
| You have managed to keep up but it's been difficult | 2 | 3 |
| You have been behind | 3 | 2 |
| You have not been able to do these activities at all | 4 | 1 |

# 28) How often does having bronchiectasis get in the way of meeting your work, household, family, or personal goals?

| Response | Score |
|-----------|-------|
| Always | 1 |
| Often | 2 |
| Sometimes | 3 |
| Never | 4 |

#### 29) Have you felt congestion (fullness) in your chest?

| Response | Score |
|-------------------|-------|
| A lot | 1 |
| A moderate amount | 2 |
| A little | 3 |
| Not at all | 4 |

#### 30) Have you been coughing during the day?

| Response | Score |
|-------------------|-------|
| A lot | 1 |
| A moderate amount | 2 |
| A little | 3 |
| Not at all | 4 |

#### 31) Have you had to cough up sputum?

| Response | Score |
|-------------------|-------|
| A lot | 1 |
| A moderate amount | 2 |
| A little | 3 |
| Not at all | 4 |

#### 32) Has your sputum been mostly:

| Response | Score | Reverse-coded Score |
|----------------------------|-------|---------------------|
| Clear | 1 | 4 |
| Clear to yellow | 2 | 3 |
| Yellowish-green | 3 | 2 |
| Brownish-dark | 4 | 1 |
| Green with traces of blood | 4 | 1 |
| Don't know | 6 | Not Scored |

# 33) Have you had shortness of breath when being more active, such as when doing housework or gardening?

| Response | Score |
|-----------|-------|
| Always | 1 |
| Often | 2 |
| Sometimes | 3 |
| Never | 4 |

#### 34) Have you been wheezing?

| Response | Score |
|-----------|-------|
| Always | 1 |
| Often | 2 |
| Sometimes | 3 |
| Never | 4 |

#### 35) Have you had chest pain?

| Response | Score |
|-----------|-------|
| Always | 1 |
| Often | 2 |
| Sometimes | 3 |
| Never | 4 |

#### 36) Have you had shortness of breath when talking?

| Response | Score |
|-----------|-------|
| Always | 1 |
| Often | 2 |
| Sometimes | 3 |
| Never | 4 |

#### 37) Have you woken up during the night because you were coughing?

| Response | Score |
|-----------|-------|
| Always | 1 |
| Often | 2 |
| Sometimes | 3 |
| Never | 4 |

If two responses are marked the worst response should be selected for scoring. This provides a conservative estimate of the response to this item.

Missing values are not imputed. If the responses are missing for more than half the items in a scale, the score for that scale should not be calculated.

Item 32 (resp32) has 5 possible answers that are scored and all other items on the questionnaire have only 4 possible answers. Possible values for resp32 are 1, 2, 3, 4, 5 (scored as 4) and 6 (not scored), whereas for other questions the possible scores are 1, 2, 3, and 4. Resp32 and eight other items are also reverse coded; because of the wording for these particular items, reverse coding is necessary to make higher scores correspond to better health outcomes. Reverse coding is conducted for resp32, and for health5, vital8, treat12, treat14, health15, role20, health24 and role27. For those items the reverse score should be used in the analysis.

The following SAS code will be used to calculate scores for the eight comains. Note that a total column score is not calculated.

#### Physical Functioning Domain

5 items: 1, 2, 3, 4, 16

if nmiss (phys1, phys2, phys3, phys4, phys16) <= 2 then
physical = (mean (phys1, phys2, phys3, phys4, phys16)-1)/3\*100;</pre>

#### • Role Functioning Domain

5 items: 17, 20, 25, 27, 28
if nmiss (role17, role20, role25, role27, role28) <= 2 then
role = (mean (role17, role20, role25, role27, role28)-1)/3\*100;</pre>

#### Vitality Domain

3 items: 6, 8, 9
if nmiss (vital6, vital8, vital9) <= 1 then
vitality = (mean (vital6, vital8, vital9)-1)/3\*100;</pre>

#### • Emotional Functioning Domain

4 items: 7, 10, 11, 23

if nmiss (emot7, emot10, emot11, emot23) <= 2 then
emotion = (mean (emot7, emot10, emot11, emot23)-1)/3\*100;</pre>

#### Social Functioning Domain

4 items: 18, 19, 22, 26
if nmiss (social18, social19, social22, social26) <= 2 then
social = (mean (social18, social19, social22, social26)-1)/3\*100;</pre>

#### • Treatment Burden Domain

3 items: 12, 13, 14

if nmiss (treat12, treat13, treat14) <= 1 then
treat = (mean (treat12, treat13, treat14)-1)/3\*100;</pre>

#### Health Perceptions Domain

4 items: 5, 15, 21, 24

if nmiss (health5, health15, health21, health24) <= 2 then
health = (mean (health5, health15, health21, health24)-1)/3\*100;</pre>

#### • Respiratory Symptoms Domain

9 items: 29, 30, 31, 32, 33, 34, 35, 36, 37

if nmiss (resp29, resp30, resp31, resp32, resp33, resp34, resp35,
resp36, resp37) <= 4 then
respirat = (mean (resp29, resp30, resp31, resp32, resp33, resp34,
resp35, resp36, resp37)-1)/3\*100;</pre>

Sponsor: Zambon S.p.A. Protocol Number: Z7224L02

# **Appendix 3: WHO-DD Preferred Terms for Antibiotics and Anti-Pseudomonal Antibiotics**

| COMMON ANTIBIOTICS WHO PT | ANTI-<br>PSEUDOMONAL |
|-------------------------------------------------|----------------------|
| ADENOMYCIN | ISECDOMONAL |
| ADICILLIN | |
| ALATROFLOXACIN | |
| AMIKACIN | Y |
| AMIKACIN SULFATE | Y |
| AMOXICILLIN | |
| AMOXICILLIN SODIUM; CLAVULANATE POTASSIUM | |
| AMOXICILLIN TRIHYDRATE | |
| AMOXICILLIN TRIHYDRATE;CLAVULANATE<br>POTASSIUM | |
| AMOXICILLIN;CLAVULANATE POTASSIUM | |
| AMOXICILLIN;CLAVULANIC ACID | |
| AMPHOTERICIN B | |
| AMPICILLIN;SULBACTAM | |
| ASPOXICILLIN | |
| ASTROMICIN | |
| AVAROFLOXACIN | |
| AVIBACTAM | Y |
| AZIDOCILLIN | |
| AZITHROMYCIN | Y |
| AZITHROMYCIN DIHYDRATE | Y |
| AZTREONAM | Y |
| BACAMPICILLIN | |
| BALOFLOXACIN | |
| BEKANAMYCIN | |
| BENZYLPENICILLIN | |
| BENZYLPENICILLIN SODIUM | |
| BRODIMOPRIM | |
| CAFROLICYCLINE | |
| CARBENICILLIN | |
| CARBOMYCIN A | |
| CARINDACILLIN | |
| CARUMONAM | |

Sponsor: Zambon S.p.A. Protocol Number: Z7224L02

| COMMON ANTIBIOTICS WHO PT | ANTI-<br>PSEUDOMONAL |
|---------------------------------------|----------------------|
| CEFACETRILE | ISECDOMONAL |
| CEFACLOR | Y |
| CEFADROXIL | Y |
| CEFALEXIN | Y |
| CEFALOGLYCIN | |
| CEFALORIDINE | |
| CEFALOTIN | |
| CEFAMANDOLE | |
| CEFAPIRIN | |
| CEFATHIAMIDINE | |
| CEFATRIZINE | Y |
| CEFAZOLIN | Y |
| CEFAZOLIN SODIUM | Y |
| CEFEPIME | Y |
| CEFIXIME | Y |
| CEFRADINE | Y |
| CEFTAZIDIME | Y |
| CEFTAZIDIME/AVIBACTAM | Y |
| CEFTOLOZANE SULFATE;TAZOBACTAM SODIUM | Y |
| CEFTOLOZANE/TAZOBACTAM | Y |
| CEFTRIAXONE | Y |
| CEFTRIAXONE SODIUM | Y |
| CEFUROXIME | Y |
| CEFUROXIME AXETIL | Y |
| CHLORAMPHENICOL | |
| CIPROFLOXACIN | Y |
| CIPROFLOXACIN HYDROCHLORIDE | Y |
| CIPROFLOXACIN LACTATE | Y |
| CLARITHROMYCIN | Y |
| CLAVULANIC ACID | |
| CLINDAMYCIN | |
| CO-AMOXICLAV | |
| COLISTIMETHATE SODIUM | Y |
| COLISTIN | Y |
| COLISTIN SULFATE | Y |
| CO-TRIMOXAZOLE | |
| DORIPENEM DOVVOYCH DIE | Y |
| DOXYCYCLINE | Y |

| | ANTI- |
|-----------------------------------------------------|-------------|
| COMMON ANTIBIOTICS WHO PT DOXYCYCLINE HYDROCHLORIDE | PSEUDOMONAL |
| ERYTHROMYCIN | Y |
| FIDAXOMICIN | Y |
| FLUCLOXACILLIN | Y |
| FOSFOMYCIN | |
| FUSIDATE SODIUM | Y |
| GENTAMICIN | Y |
| IMIPENEM | Y |
| IMIPENEM/CILASTATIN | Y |
| LEVOFLOXACIN | Y |
| LINCOMYCIN HYDROCHLORIDE | |
| MEROPENEM | Y |
| MEROPENEM TRIHYDRATE | Y |
| METHENAMINE | |
| METHENAMINE HIPPURATE | |
| METRONIDAZOLE | |
| MOXIFLOXACIN | Y |
| MOXIFLOXACIN HYDROCHLORIDE | Y |
| NITROFURANTOIN | |
| OFLOXACIN | |
| PIPERACILLIN | Y |
| PIPERACILLIN SODIUM;TAZOBACTAM SODIUM | Y |
| PIPERACILLIN;TAZOBACTAM | Y |
| POLYMYXIN B | |
| ROXITHROMYCIN | Y |
| SULFAMETHOXAZOLE | |
| SULFAMETHOXAZOLE;TRIMETHOPRIM | |
| SULTAMICILLIN | |
| TAZOBACTAM | Y |
| TOBRAMYCIN | Y |
| TOBRAMYCIN SULFATE | Y |
| TRIMETHOPRIM | |

### Z7224L02\_SAP\_v4\_FINAL\_08.02.2022

Final Audit Report 2022-04-08

Created: 2022-04-08

By: PPD

Status: Signed

Transaction ID: CBJCHBCAABAAsB5gLhyJIPIPCdlPaFGyuXz9MfmG2OPL

### "Z7224L02\_SAP\_v4\_FINAL\_08.02.2022" History

Document created by PPD

2022-04-08 - 14:06:31 GMT- IP address: 147.161.167.17

Document emailed to PPD

2022-04-08 - 14:10:32 GMT

Document emailed to PPD for signature

2022-04-08 - 14:10:32 GMT

Document emailed to PPD for signature

2022-04-08 - 14:10:32 GMT

✓ PPD verified identity with Adobe Acrobat Sign authentication

for signature

2022-04-08 - 14:11:38 GMT

Signature Date: 2022-04-08 - 14:11:38 GMT - Time Source: server- IP address: 147.161.167.17

🖰 Email viewed by PPD

2022-04-08 - 14:15:33 GMT- IP address: 104.47.5.254

✓ PPD verified identity with Adobe Acrobat Sign authentication

2022-04-08 - 14:30:50 GMT

Signature Date: 2022-04-08 - 14:30:50 GMT - Time Source: server- IP address: 93.34.125.117

Email viewed by PPD

2022-04-08 - 16:21:37 GMT- IP address: 104.47.4.254

✓ PPD verified identity with Adobe Acrobat Sign authentication

2022-04-08 - 16:26:01 GMT



Powered by Adobe Acrobat Sign Document e-signed by PPD

Signature Date: 2022-04-08 - 16:26:01 GMT - Time Source: server- IP address: 109.154.73.148

Agreement completed.

2022-04-08 - 16:26:01 GMT



Powered by Adobe Acrobat Sign